A RANDOMIZED, CONTROLLED, OPEN-LABEL SHORT-TERM STUDY TO EVALUATE CHANGES IN EXPOSURE TO HARMFUL AND POTENTIALLY HARMFUL CONSTITUENTS IN ADULT SMOKERS WHO PARTIALLY OR COMPLETELY SWITCH TO VERVE® PRODUCTS (DISCS OR CHEWS) IN A CLINICAL SETTING

NCT03692078

06AUG2018



## Statistical Analysis Plan

A RANDOMIZED, CONTROLLED, OPEN-LABEL SHORT-TERM STUDY TO EVALUATE CHANGES IN EXPOSURE TO HARMFUL AND POTENTIALLY HARMFUL CONSTITUENTS IN ADULT SMOKERS WHO PARTIALLY OR COMPLETELY SWITCH TO VERVE® PRODUCTS (DISCS OR CHEWS) IN A CLINICAL SETTING

Protocol No. ALCS-RDS-18-04-VRV Celerion Project CA24563 Final Version 1.2 Date: 06 August 2018

Final Protocol Date: 30 March, 2018 Final Protocol Amendment 1 Date: 25 May 2018

> Altria Client Services LLC 601 E. Jackson Street Richmond, Virginia 23219

Celerion 621 Rose Street Lincoln, Nebraska 68502

## Statistical Analysis Plan Signature Page

Altria Client Services LLC 601 E. Jackson Street Richmond, Virginia 23219

Protocol: ALCS-RDS-18-04-VRV

Title: A RANDOMIZED, CONTROLLED, OPEN-LABEL SHORT-TERM STUDY TO EVALUATE CHANGES IN EXPOSURE TO HARMFUL AND POTENTIALLY HARMFUL CONSTITUENTS IN ADULT SMOKERS WHO PARTIALLY OR COMPLETELY SWITCH TO VERVE® PRODUCTS (DISCS OR CHEWS) IN A CLINICAL SETTING

Issue Date: 06 August 2018



# **TABLE OF CONTENTS**

| 1. | INT | RODUC | CTION | | | 7 |
|---|---|---|---|---|---|---|
| 2. | STU | DY PU | RPOSE, H | <b>IYPOTHES</b> | IS, OBJECTIVES AND ENDPOINTS | 7 |
| | 2.1 | Study | Purpose | | | 7 |
| | 2.2 | | _ | | | |
| | 2.3 | Objec | tives | | | 7 |
| | | 2.3.1 | Primary | Objective | | 7 |
| | | 2.3.2 | Secondar | ry Objective | s | 7 |
| | 2.4 | Outco | me Variab | les | | 8 |
| 3. | STU | DY DE | SIGN | | | 9 |
| 4. | SAN | <b>IPLE S</b> | IZE ESTIN | MATION | | 12 |
| 5. | | | | | | |
| 6. | STU | DY GR | OUP ANI | O PRODUC | T DESCRIPTIONS | 13 |
| 7. | BIO | MARK | ER ASSES | SSMENT A | ND ANALYSIS | 14 |
| | 7.1 | Bioma | | | on and Measurements | |
| | | 7.1.1 | Urine Bi | | Exposure (BOE) | |
| | | | 7.1.1.1 | | E Sample Collection | |
| | | | 7.1.1.2 | | cal Method | |
| | | | 7.1.1.3 | Urine Bion | narker Analysis Variables | |
| | | | | 7.1.1.3.1 | Urine Nicotine Equivalents | 15 |
| | | | | 7.1.1.3.2 | Urine Biomarkers Adjusted for Urine | |
| | | | | | Creatinine | |
| | | | | 7.1.1.3.3 | Urine Biomarker Change From Baseline | |
| | | | | 7.1.1.3.4 | Urine Mutagenicity | |
| | | 7.1.2 | | | Exposure | |
| | | | 7.1.2.1 | | E Sample Collection | |
| | | | 7.1.2.2 | • | cal Method | |
| | | 710 | 7.1.2.3 | | marker Analysis Variables | |
| | | 7.1.3 | | | illection and Analysis Variables | |
| | | | 7.1.3.1 | | ection | |
| | | 714 | 7.1.3.2 | - | Variables | |
| | | 7.1.4 | 7 1 4 1 | | ation | |
| | | | 7.1.4.1 | | ection | |
| | 7.2 | Doto S | | | Variablestion | |
| | 1.2 | 7.2.1 | • | | ary | |
| | | 7.2.1 | _ | - | ary | |
| | | 7.2.2 | _ | | | |
| | | 7.2.3 | | | | |
| | | 7.2.4 | | | | |
| | | , | ~ ~~~ | | | |

| | 7.3 Statistical Analyses | | | | 22 |
|---|---|---|---|---|---|
| | • | | | Endpoint Analysis | |
| | | | 7.3.1.1 | | |
| | | | 7.3.1.2 | Dealing with non-normality | |
| | <ul><li>7.3.2 Secondary Endpoint Analysis</li><li>7.3.3 Subjective Effects</li></ul> | | | | |
| | | 7.3.4 | - | ity Analysis | |
| | | | 7.3.4.1 | Analysis Variables for Sensitivity Analysis | 24 |
| | | | 7.3.4.2 | Handling of Missing Data | |
| | | | 7.3.4.3 | | |
| | | | 7.3.4.4 | Handling BLQ values | |
| 8. | SAFETY | | | | |
| | 8.1 Subject Disposition | | | | 26 |
| | 8.2 Adverse Events. | | | | |
| | 8.3 Clinical Laboratory | | | | |
| | 8.4 Vital Signs | | | | |
| | 8.5 ECG | | | | |
| | 8.6 Concomitant Medications | | | | |
| | 8.7 Physical Examination. | | | | |
| 9. | SUN | _ | | ANGES FROM PROTOCOL-PLANNED ANALYSIS | |
| 10. | SUM | <b>IMARY</b> | TABLES | S AND FIGURES | 28 |
| 12. | TABLE SHELLS | | | | 40 |
| 13. | LISTING SHELLS | | | | |
| 14. | FIGURE SHELLS 12 | | | | |
| 15. | REFERENCES | | | | 130 |

#### ABBREVIATIONS AND DEFINITIONS

1-OHP 1-hydroxypyrene 1-OHPhe 1-OH-Phenanthrene 2-AN 2-aminonaphthalene

2-HPMA 2-hydroxypropyl-mercapturic acid 2-MHBMA 2-hydroxybutenyl-mercapturic acid

2-OHFle 2 OH-Fluorene

3-HMPMA 3-hydroxy-1-methylpropylmercapturic acid

3-HPMA 3-hydroxypropylmercapturic acid

4-ABP 4-aminobiphenyl

AAMA N-acetyl-S-(2-carbamoylethyl)-l-cysteine

AE adverse event

AIC Akaike information criterion ALCS Altria Client Services LLC ANCOVA analysis of covariance

BLQ below the limit of quantitation

BMI body mass index

BOE biomarker of exposure BOPH biomarker of potential harm CEMA 2-cyanoethylmercapturic acid

confidence interval CI carbon monoxide CO COHb carboxyhemoglobin cigarettes per day CPD **CSR** clinical study report coefficient of variation CV**ECG** electrocardiogram end-of-study EOS

FTCD Fagerström Test for Cigarette Dependence

GAMA N-acetyl-S-(2-carbamoyl-2-hydroxyethyl)-l-cysteine

HEMA 2-hydroxyethyl mercapturic acid

HPHC harmful and potentially harmful constituents

ICF informed consent form

ICH International Conference on Harmonization

ITT intent to treat kg kilogram(s)

LC-MS liquid chromatography–mass spectrometry

LLOQ lower limit of quantitation LLC limited liability company

m meter(s)

mCEQ modified Cigarette Evaluation Questionnaire MedDRA Medical Dictionary for Regulatory Activities

mg milligram(s)

mITT modified intent to treat

mL milliliter(s)

MMRM mixed model for repeated measures N, n sample size, number of observations

NE nicotine Equivalents

ng nanograms

NNAL 4-(methylnitrosamino)-1-(3-pyridyl)-1-butanol

NNN N-nitrosonornicotine

OB own brand

OTDN oral tobacco-derived nicotine

pg pictogram
PP per-protocol
Q1 first quartile
Q3 third quartile

SAE serious adverse event SAP statistical analysis plan SD standard deviation

SEM standard error of the mean S-PMA S-phenyl mercapturic acid

μg microgram

VPD VERVE® product(s) per day

WHO-DD World Health Organization Drug Dictionary

#### 1. INTRODUCTION

The following Statistical Analysis Plan (SAP) provides the framework for the summarization of the data from this study. The analysis plan may change due to unforeseen circumstances. Any changes made after locking of the database will be documented in the Clinical Study Report (CSR).

Any additional analyses not addressed within this SAP and/or driven by the data, or requested by Altria Client Services LLC, will be considered out of scope and must be approved, by Altria Client Services LLC, and must be described in the CSR.

### 2. STUDY PURPOSE, HYPOTHESIS, OBJECTIVES AND ENDPOINTS

## 2.1 Study Purpose

The purpose of this study is to evaluate changes in exposure to selected harmful and potentially harmful constituents (HPHC) by measuring biomarkers in adult smokers who partially or completely switch from smoking to oral tobacco-derived nicotine (OTDN) products VERVE® Chews or VERVE® Discs use compared to those who continue exclusively smoking cigarettes or stop using all tobacco products.

## 2.2 Hypothesis:

Reducing daily cigarette consumption by at least 50% and using VERVE $^{\text{@}}$  products will result in a statistically significant reduction in 24-hour urinary total 4-(methylnitrosamino)-1-(3-pyridyl)-1-butanol (NNAL) on Day 7 compared to continued cigarette smoking.

## 2.3 Objectives

### 2.3.1 Primary Objective

The primary objective is to:

To compare 24-hour urinary total NNAL in adult smokers who reduce cigarette consumption by at least 50% with supplementary (dual) usage of VERVE® Chews or VERVE® Discs to those who continue to smoke cigarettes for 7 days.

### 2.3.2 Secondary Objectives

The secondary objectives are to:

1. To compare biomarkers of exposure (total N-nitrosonornicotine [NNN], nicotine equivalents [NE], 2-aminonaphthalene [2-AN], 4-aminobiphenyl [4-ABP], 2-hydroxyethyl mercapturic acid [HEMA], 2-cyanoethylmercapturic acid [CEMA], S-phenyl mercapturic acid [S-PMA], 3-hydroxy-1-methylpropylmercapturic acid [3-HMPMA], 3-hydroxypropylmercapturic acid [3-HPMA], 2-hydroxypropyl-mercapturic acid [2-HPMA], N-acetyl-S-(2-carbamoylethyl)-1-cysteine [AAMA], N-acetyl-S-(2-carbamoyl-2-hydroxyethyl)-1-cysteine [GAMA], 2-hydroxybutenyl-mercapturic acid [2-MHBMA], 2-OH-

- Fluorene [2-OHFle], 2-Naphthol,1-OH-Phenanthrene [1-OHPhe], urine mutagenicity, 1-hydroxypyrene [1-OHP], and carboxyhemoglobin [COHb]) in adult smokers who reduce cigarette consumption by at least 50% with supplementary (dual) usage of VERVE® Chews or VERVE® Discs to those who continue to smoke cigarettes for 5 and 7 days.
- 2. To compare 24-hour urinary total NNAL in adult smokers who reduce cigarette consumption by at least 50% with supplementary (dual) usage of VERVE® Chews or VERVE® Discs to those who continue to smoke cigarettes for 5 days.
- 3. To compare biomarkers of exposure (total NNAL, total NNN, NE, 2-AN, 4-ABP, HEMA, CEMA, S-PMA, 3-HMPMA, 3-HPMA, 2-HPMA, AAMA, GAMA, 2-MHBMA, 2-OHFle, 2-Naphthol, 1-OHPhe, urine mutagenicity, 1-OHP and COHb) in adult smokers who reduce cigarette consumption by at least 50% with supplementary (dual) usage of VERVE® Chews or VERVE® Discs to those who cease from all tobacco use for 5 and 7 days.
- 4. To compare biomarkers of exposure (total NNAL, total NNN, NE, 2-AN, 4-ABP, HEMA, CEMA, S-PMA, 3-HMPMA, 3-HPMA, 2-HPMA, AAMA, GAMA, 2-MHBMA, 2-OHFle, 2-Naphthol, 1-OHPhe, urine mutagenicity, 1-OHP and COHb) in adult smokers who completely switch to VERVE® Chews or VERVE® Discs to those who continue to smoke cigarettes for 5 and 7 days.
- 5. To compare biomarkers of exposure (total NNAL, total NNN, NE, 2-AN, 4-ABP, HEMA, CEMA, S-PMA, 3-HMPMA, 3-HPMA, 2-HPMA, AAMA, GAMA, 2-MHBMA, 2-OHFle, 2-Naphthol, 1-OHPhe, urine mutagenicity, 1-OHP and COHb) in adult smokers who completely switch to VERVE® usage to those who cease from all tobacco use for 5 and 7 days.
- 6. To compare subjective effects (Questionnaire of Smoking Urges Brief [QSU-Brief] total score, responses to modified cigarette evaluation questionnaire [mCEQ] and the Use the Product Again questionnaire) among subjects who continue to smoke cigarettes, subjects with dual usage of VERVE® Chews or VERVE® Discs and cigarettes, subjects with complete switch to VERVE® Chews or VERVE® Discs, and subjects who cease from all tobacco use for 1, 5 and 7 days.
- 7. To characterize product use behaviors (such as: number of cigarettes per day [CPD], number of VERVE® use per day [VPD], average and total duration of VERVE® use each day).

#### 2.4 Outcome Variables

#### **Primary**

The primary outcome variable is:

• 24-hour total urinary NNAL (ng/24 hours) excreted on Day 7.

### Secondary

The secondary outcome variables are:

- 24-hour urinary total total NNN, NE, 2-AN, 4-ABP, HEMA, CEMA, S-PMA, 3-HMPMA, 3-HPMA, 2-HPMA, AAMA, GAMA, 2-MHBMA, 2-OHFle, 2-Naphthol, 1-OHPhe, mutagenicity, and 1-OHP excreted on Day 5 and Day 7.
- 24-hour urinary total NNAL excreted on Day 5.
- COHb on Day 5 and Day 7.
- QSU-Brief responses and factor scores on Day 1, Day 5, and Day 7.
- Responses to the appropriate mCEQ on Day 1, Day 5, and Day 7.
- Responses to the appropriate Use the Product Again questionaire on Day 7.
- Product use behavior daily from Day 1 to Day 7 (i.e., CPD, VPD, and the average and total duration of VERVE® product use each day).

## **Clinical Safety**

- AEs and SAEs
- ECG, vital signs, clinical chemistry, urinalysis, and hematology

#### 3. STUDY DESIGN

This is an open label, randomized, 6 parallel-group clinical study evaluating changes in exposure to selected HPHCs, subjective effects, and product use behavior in adult smokers who are randomly assigned to continue smoking, partially or completely switch to VERVE<sup>®</sup> Chews or VERVE<sup>®</sup> Discs products, or stop using all tobacco products for 7 days.

The overall design of the study is shown in Figure 1.

Figure 1: Overall Study Design



**Study Products:** 

Product A: Subject's own brand (OB) Cigarette (Reference Product)

Product B: Oral tobacco-derived nicotine chews marketed as VERVE®

Discs Blue Mint (~1.5 mg nicotine/piece) (Test Product)

Product C: Oral tobacco-derived nicotine chews marketed as VERVE®

Discs Green Mint (~1.5 mg nicotine/piece) (Test Product)

Product D: Oral tobacco-derived nicotine chews marketed as VERVE®

Chews Blue Mint (~1.5 mg nicotine/piece) (Test Product)

Product E: Oral tobacco-derived nicotine chews marketed as VERVE®

Chews Green Mint (~1.5 mg nicotine/piece) (Test Product)

Approximately 210 healthy adult male and female (no more than 60% of either gender) self-affirmed combustible cigarette smokers, 21 - 65 years of age, inclusive (determined at Screening), willing to abstain from smoking and use all four VERVE® products, and who fulfill all inclusion criteria and none of the exclusion criteria will be enrolled. All subjects must have an average daily consumption of at least 10 but no more than 30 factory manufactured combustible cigarettes for at least 12 months prior to Screening. Use of other types of tobacco- or nicotine-containing products will not be permitted within 1 week prior to Check-in.

Subjects, who meet all inclusion criteria and none of the exclusion criteria, will check-in to the clinic on Day -3 at a time determined by the clinic. After check-in, subjects will engage in a brief product trial with each flavor of VERVE® Chews (two flavors: blue mint and green mint) and VERVE® Discs (two flavors: blue mint and green mint). This trial period will involve *ad libitum* use for 10 minutes each to allow subjects to become accustomed to using the products. The trial of each flavor of VERVE® Chews or VERVE® Discs product will be separated by approximately 30 minutes (from the start of each product trial). Subjects who are unwilling to use and/or cannot tolerate all four VERVE® products will not continue in the study.

Following completion of the VERVE® product trial on Day -3, subjects will continue to smoke their OB cigarettes through 23:00 on Day -3 and from 07:00 to 23:00 on Days -2 and -1. Baseline cigarette consumption for each subject will be determined by the average number of cigarettes smoked (CPD) on Day -2 and Day -1 and will be used to calculate the CPD allowed for each subject in Group 2 or Group 3, according to their assigned randomization group, for the remainder of the study. Other baseline study events will include 24-hour urine collections for biomarkers of exposure (total NNAL, total NNN, NE, 2-AN, 4-ABP, HEMA, CEMA, S-PMA, 3-HMPMA, 3-HPMA, 2-HPMA, AAMA, GAMA, 2-MHBMA, 2-OHFle, 2-Naphthol, 1-OHPhe, mutagenicity, and 1-OHP), blood sampling for COHb, and administration of the QSU-Brief and the appropriate mCEQ questionnaire on Day -1.

On Day 1, subjects will be randomized into one of the following Groups:

• GROUP 1 (n = 40): Continue Smoking

Subjects will be asked to continue smoking their OB cigarettes ad libitum for 7 days.

• GROUP 2 (n = 40): VERVE® Discs Dual Use

Subjects will reduce their normal daily cigarette consumption by at least 50% of their baseline CPD and use at least 3 VERVE® Discs per day for 7 days.

• GROUP 3 (n = 40): VERVE<sup>®</sup> Chews Dual Use

Subjects will reduce their normal daily cigarette consumption by at least 50% of their baseline CPD and use at least 3 VERVE® Chews per day for 7 days.

- GROUP 4 (n = 30): VERVE<sup>®</sup> Discs Exclusive Use Subjects will completely switch to exclusive use of VERVE<sup>®</sup> Discs, using at least 3 discs per day for 7 days.
- GROUP 5 (n = 30): VERVE<sup>®</sup> Chews Exclusive Use Subjects will completely switch to exclusive use of VERVE<sup>®</sup> Chews, using at least 3 chews per day for 7 days.
- GROUP 6 (n = 30): Tobacco Cessation Subjects will completely stop all tobacco product usage for 7 days.

Subjects will be randomized into each Group on Day 1 based on gender and CPD.

Subjects will begin using the assigned study products or completely stop using tobacco products on the morning of Day 1 and continue through discharge according to the randomization.

On each study day (Days 1 - 7), subjects in Group 1 will be allowed to smoke their OB cigarettes *ad libitum* (i.e., no restriction on the duration of use or the number of cigarettes per day) from 07:00 through 23:00. Subjects will be allowed to smoke upon request to the clinic staff but will only be allowed 1 cigarette at a time and will be instructed to return each cigarette butt upon completion.

On each study day (Days 1 - 7), subjects in Group 2 and Group 3 will smoke no more than 50% of their baseline CPD and will use the assigned VERVE® product *ad libitum* (i.e., no restrictions on the number of VERVE® products used at once, the number of VERVE® products used per day, or the duration of use) except for 3 specific VERVE® products use opportunities at approximately 11:00, 15:00, and 19:00 each day during which subjects will be asked to keep the assigned VERVE® product in their mouth for at least 10 minutes. Subjects will be allowed to smoke upon request to the clinic staff but will only be allowed 1 cigarette at a time and will be instructed to return each cigarette butt upon completion. Subjects will be allowed to use the VERVE® product upon request [more then 1 permitted at a time, but all returned before more are dispensed] and they will be instructed to return each used VERVE® product upon completion.

On each study day (Days 1 - 7), subjects in Group 4 and Group 5 will use the assigned VERVE® product *ad libitum* (i.e., no restrictions on the number of VERVE® products used at once, the number of VERVE® products used per day, or the duration of use) except for 3 specific VERVE® products use opportunities at approximately

11:00, 15:00, and 19:00 each day during which subjects will be asked to keep the assigned VERVE® product in their mouth for at least 10 minutes. Subjects will be allowed to use the VERVE® product upon request [more then 1 permitted at a time, but all returned before more are dispensed] and they will be instructed to return each used VERVE® product upon completion.

On each study day (Days 1 - 7), subjects in Group 6 will completely stop cigarette use and they will not be allowed to smoke or use  $VERVE^{®}$  products.

All product use (CPD, VPD, and VERVE® product use duration, [i.e., time of VERVE® product placement in the subjects' mouth, and time it was removed from the subjects' mouth], as appropriate) will be determined to assess product use behavior.

Study events will include 24-hour urine collections for biomarkers of exposure (total NNAL, total NNN, NE, 2-AN, 4-ABP, HEMA, CEMA, S-PMA, 3-HMPMA, 3-HPMA, 2-HPMA, AAMA, GAMA, 2-MHBMA, 2-OHFle, 2-Naphthol, 1-OHPhe, mutagenicity, and 1-OHP) and blood sample collection for COHb assessment. Urine creatinine will be measured in each 24-hour collection and will be used to adjust the concentration values of urine biomarkers. Each 24-hour urine collection (Day -1, Day 5 and Day 7) will be from approximately (± 30 minutes) 07:00 on the scheduled day to approximately 07:00 the following day. The 24-hour urine collection begins on each scheduled day after the first morning void and any void prior to 07:00, and finishes the following morning with the last void collected at approximately 07:00 (including first morning void). Subjects will be specifically instructed to collect all urine voided, and any missed collection during the 24-hour interval will be documented as a deviation.

Subjects will also complete in the moment subjective effects questionnaires, which include QSU-Brief (Protocol Appendix 2), Modified Cigarette Evaluation Questionnaire (mCEQ-C & mCEQ-V; Protocol Appendix 3), and Use the Product Again questionnaire (UPA-C & UPA-V; Protocol Appendix 4). Details for subject effect data collection is in Section 7.1.4.1.

### 4. SAMPLE SIZE ESTIMATION

This study is designed to evaluate changes in exposure to selected HPHC when adult smokers partially or completely switch to oral tobacco-derived nicotine VERVE® Chews or VERVE® Discs compared to those who continue smoking cigarettes or stop using all tobacco products. Assuming a similar effect size for the new study as for the previous ALCS study (ToPP4ST\_1011\_07) between the continued cigarette smoking group and each of the two dual usage groups ( $\geq$ 50% CPD reduction with VERVE® DISCS or VERVE® CHEWS), a two-sided t test, 85% power and an  $\alpha$  =0.025 Type I error rate to account for the multiplicity adjustment for the two comparisons, 35 subjects are needed to complete for the continue cigarette smoking group and the dual usage groups. We expect that the effect will be larger in the VERVE® only and smoking cessation groups, so 25 subjects are needed to complete in these groups.

#### 5. ANALYSIS POPULATIONS

## **Safety Analysis Dataset:**

All subjects who used any study products (including subjects randomized to Group 6).

## **Modified Intent-to-Treat (mITT) Dataset:**

All randomized subjects who used at least one study product after randomization (except Group 6) and have a valid baseline and at least one post-baseline biomarker measure of any one biomarker.

## Per-Protocol (PP) Dataset:

A subset of the mITT dataset and includes subjects who completed the study without important (or major) protocol deviations that are considered to impact data integrity (e.g., non adherence to study group assignment).

If it is determined that a subject was pregnant during the study, all of the pregnant subject's data will be reported, but will be excluded from summarization and statistical analyses.

## 6. STUDY GROUP AND PRODUCT DESCRIPTIONS

The following products will be tested in this study:

- Product A: Subject's OB Cigarette (Reference Product)
- Product B: Oral tobacco-derived nicotine chews marketed as VERVE® Discs Blue Mint (~1.5 mg nicotine/piece) (Test Product)
- Product C: Oral tobacco-derived nicotine chews marketed as VERVE® Discs Green Mint (~1.5 mg nicotine/piece) (Test Product)
- Product D: Oral tobacco-derived nicotine chews marketed as VERVE® Chews Blue Mint (~1.5 mg nicotine/piece) (Test Product)
- Product E: Oral tobacco-derived nicotine chews marketed as VERVE® Chews Green Mint (~1.5 mg nicotine/piece) (Test Product)

The following groups will be tested in this study and the group descriptions will be used in the footnotes for listings, tables, and figures:

- **GROUP 1: Continue Smoking**
- GROUP 2: VERVE® Discs Dual Use
- GROUP 3: VERVE® Chews Dual Use
- GROUP 4: VERVE® Discs Exclusive Use
- GROUP 5: VERVE® Chews Exclusive Use
- **GROUP 6: Tobacco Cessation**

Study groups will be referred to in the text as: Continue Smoking Group, VERVE<sup>®</sup> Discs Dual Use Group, VERVE<sup>®</sup> Chews Dual Use Group, VERVE<sup>®</sup> Discs Exclusive Use Group, VERVE<sup>®</sup> Chews Exclusive Use Group, and Tobacco Cessation Group.

### 7. BIOMARKER ASSESSMENT AND ANALYSIS

## 7.1 Biomarkers Sample Collection and Measurements

## 7.1.1 Urine Biomarkers of Exposure (BOE)

# 7.1.1.1 Urine BOE Sample Collection

24-hour urine collections for biomarkers of exposure (total NNAL, total NNN, NE, 2-AN, 4-ABP, HEMA, CEMA, S-PMA, 3-HMPMA, 3-HPMA, 2-HPMA, AAMA, GAMA, 2-MHBMA, 2-OHFle, 2-Naphthol, 1-OHPhe, mutagenicity, and 1-OHP) will be performed on Days -1, 5, and 7. Urine creatinine will be measured in each 24-hour collection and will be used to adjust the concentration values of urine biomarkers. Each 24-hour urine collection will be from approximately (± 30 minutes) 07:00 on the scheduled day to approximately 07:00 the following day. The 24-hour urine collection begins on each scheduled day after the first morning void and any void prior to 07:00, and finishes the following morning with the last void collected at approximately 07:00 (including first morning void). Subjects will be specifically instructed to collect all urine voided, and any missed collection during the 24-hour interval will be documented as a deviation.

## 7.1.1.2 Bioanalytical Method

Urine aliquots for NE will be shipped to Celerion Bioanalytical Services for analysis. These samples will be analyzed using validated LC-MS/MS analytical methods.

Aliquots for creatinine will be shipped to the Celerion Clinical Laboratory for analysis.

Urine aliquots for NNAL, NNN, 2-AN, 4-ABP, HEMA, CEMA, S-PMA, 3-HMPMA, 3-HPMA, 2-HPMA, AAMA, GAMA, 2-MHBMA, 2-OHFle, 2-Naphthol, 1-OHPhe, and 1-OHP will be shipped to ABF for analysis.

Mutagenicity testing will be done by Labstat.

## 7.1.1.3 Urine Biomarker Analysis Variables

The following variables will be determined for each urine biomarker except mutagenicity testing.

- Measured concentration
- Total biomarker mass excreted per 24 hours (primary analysis variable)
- Total mass excreted per 24 hours absolute change from Baseline
- Total mass excreted per 24 hours percent change from Baseline
- Measured concentration adjusted for urine creatinine

Urine biomarker concentration values reported as below the limit of quantitation (BLQ) will be set to one-half of the limit of quantitation prior to calculating the 24-hour mass excreted. Total urine weight (g) will be collected during the study and converted to urine volume using the assumed density of 1 gram (g) equals 1 milliliter (mL).

Creatinine-adjusted concentrations will be calculated as shown in Section 7.1.1.3.2. Absolute and percent change from baseline will be calculated as shown in Section 7.1.1.3.3.

## 7.1.1.3.1 Urine Nicotine Equivalents

NE will be calculated as the molar sum of nicotine and 5 major nicotine metabolites excreted in urine over 24 hours. Values of individual components reported as below the limit of quantitation will be set to one-half of the limit of quantitation prior use in the calculation below.

The concentration of each metabolite will first be multiplied by the 24-hour urine volume to obtain the total amount excreted in 24 hours, then divided by the molecular weight of the metabolite to obtain the total amount of each in moles. The sum in moles will then be converted to mass of NE by multiplying by the molecular weight of nicotine.

| Nicotine (mg/24h) | = | nicotine concentration [ng/mL] $\times$ 24h urine volume [mL] $\div$ 1000 000 |
|---|---|---|
| Nicotine-glucuronide (mg/24h) | = | nicotine glucuronide concentration [ng/mL] × 24h urine volume [mL] ÷ 1000 000 |
| Cotinine (mg/24 hours) | = | cotinine concentration [ng/mL] $\times$ 24h urine volume [mL] $\div$ 1000 000 |
| Cotinine-glucuronide (mg/24h) | = | cotinine glucuronide concentration [ng/mL] × 24h urine volume [mL] ÷ 1000 000 |
| Trans-3'-hydroxycotinine (mg/24h) | = | trans-3'-hydroxycotinine concentration [ng/mL] × 24h urine volume [mL] ÷ 1000 000 |
| Trans-3'-hydroxycotinine-glucuronide (mg/24h) | = | trans-3'-hydroxycotinine glucuronide concentration [ng/mL] × 24h urine volume [mL] ÷ 1000 000 |

Nicotine equivalents (mg/24 hours)

= (nicotine [mg/24h]/162.23 [mg/mmol] + nicotine-gluc [mg/24h]/338.36 [mg/mmol] + cotinine [mg/24h]/176.22 [mg/mmol] + cotinine-gluc [mg/24h]/352.34 [mg/mmol] + trans-3'-hydroxycotinine [mg/24h]/192.22 [mg/mmol] + trans-3'-hydroxycotinine-gluc [mg/24h]/368.34 [mg/mmol]) x 162.23 (mg/mmol)

## 7.1.1.3.2 Urine Biomarkers Adjusted for Urine Creatinine

Urine creatinine concentration will also be measured in urine collections and will be used to adjust the concentration values of urine biomarkers except mutagenicity as follows:

### **Nicotine Equivalents**

Nicotine equivalents (mg/g creatinine) =  $\frac{\text{nicotine equivalents (µg/mL) x 100}}{\text{creatinine (mg/dL)}}$ 

## **Other Urine Biomarkers**

Urine biomarker (unit2/g creatinine) = <u>urine biomarker (unit1/mL) x 100</u> creatinine (mg/dL) Where: if unit1 = pg, then unit2 = ng and if unit1 = ng, then unit2 =  $\mu$ g

## 7.1.1.3.3 Urine Biomarker Change From Baseline

Urine biomarker change from baseline will be calculated as follows, where Baseline = Day -1:

Absolute change from baseline = Post Randomization Value – Baseline Value

Percent change from baseline (%) = (Post Randomization Value – Baseline Value) / Baseline Value x 100 %

## 7.1.1.3.4 Urine Mutagenicity

Urine mutagenicity will be analyzed and reported by Labstat.

250 mL urine sample will be concentrated to 1 mL and used for urine mutagenicity testing. The measurement results will be reported as revertants/ $\mu$ L. The urine mutagenicity count in the 24 hour urine will be calculated as follow:

Urine mutagenicity (revertants/250 mL) = Urine mutagenicity (revertants/ $\mu$ L) x 1000

Note: the coefficient 1000 is for 1 mL = 1000  $\mu$ L. If the volume after concentration is X mL, the coefficient will be X\*1000.

Urine mutagenicity (revertants/24 hour) = Urine mutagenicity (revertants/250 mL) x urine volume/250

Note: the coefficient 250 is the volume of urine sample used for mutagenicity test. If the sample volume is XXX mL, the coefficient will be XXX.

## 7.1.2 Blood Biomarkers of Exposure

## 7.1.2.1 Blood BOE Sample Collection

The blood sample for COHb will be collected 15 minutes to 45 minutes following the start of subject's in the moment subjective questionnaires (QSU-Brief, mCEQ, and Use Product Again, as appropriate) at 21:30 (±30 minutes) on Days -1, 5, and 7. Subjects will abstain from product use, as appropriate, for at least 15 minutes prior to blood draw for COHb.

## 7.1.2.2 Bioanalytical Method

Blood samples for COHb saturation will be shipped to the Celerion Clinical Laboratory for analysis. COHb saturation will be determined using a validated spectrophotometric method at the Celerion Clinical Laboratory, Lincoln, Nebraska.

## 7.1.2.3 Blood Biomarker Analysis Variables

The following variables will be determined for blood COHb.

- Measured saturation (%) (primary analysis variable)
- Measured saturation (%) absolute change from Baseline
- Measured saturation (%) percent change from Baseline

Values reported as below the limit of quantitation (BLQ) will be set to one-half of the limit of quantitation for summarization and statistical analysis.

Absolute and percent change from baseline will be calculated as shown in Section 7.1.1.3.3.

## 7.1.3 Product Use Data Collection and Analysis Variables

#### 7.1.3.1 Data Collection

Subjects will use the assigned products or be abstinent, as per randomization. All subjects (except Group 6) will use the assigned study product ad libitum (except

during meals and study procedures, as appropriate) from 07:00 through 23:00. Subjects in Group 2 and Group 3 will smoke no more than 50% of their baseline CPD and will use assigned VERVE® product ad libitum except for 3 specific VERVE® product use opportunities at 11:00, 15:00, and 19:00 each day during which subjects will be asked to keep VERVE® product in their mouth for at least 10 minutes. Subjects in Group 4 and Group 5 will only use the assigned VERVE® product ad libitum except for 3 specific VERVE® product use opportunities at 11:00, 15:00, and 19:00 each day during which subjects will be asked to keep assigned VERVE® product in their mouth for at least 10 minutes. Subjects will abstain from any product use from the start of the subjective effects questionnaires administration scheduled for 21:30 (±30 minutes) until after the COHb sample has been collected on Days -1, 5, and 7.

The number of each product used per day (CPD and VPD, as appropriate) will be counted for each cigarette or VERVE® product used during each day in a product use period. The total duration of each VERVE® product will be the sum of product use durations during each day in a product use period. The average duration of each VERVE® product will be the average of product use durations used per use each day in a product use period.

## 7.1.3.2 Analysis Variables

- number of each product used per day (CPD and VPD, as appropriate)
- average duration of VERVE® product used per use each day
- total duration of VERVE® product used per day

### 7.1.4 Subjective Effect

### 7.1.4.1 Data Collection

Subjects will also complete in the moment subjective effects questionnaires, which include:

- QSU-Brief (Protocol Appendix 2) All subjects will complete the QSU-Brief on Days -1, 1, 5, and 7 in the morning at 07:00 (± 30 minutes) before product use, as appropriate, and at 21:30 (± 30 minutes).
- Modified Cigarette Evaluation Questionnaire (mCEQ-C or mCEQ-V; Protocol Appendix 3) the appropriate mCEQ will be administered at 21:30 (± 30 minutes). All subjects will complete the mCEQ-C on Day -1. Subjects in Group 1 will also complete the mCEQ-C on Days 1, 5, and 7. Subjects in Groups 2 and 3 will complete both of the mCEQ-C and mCEQ-V on Days 1, 5, and 7. Subjects in Groups 4 and 5 will complete mCEQ-V on Days 1, 5, and 7.
- Use the Product Again questionnaire (Protocol Appendix 4) Subjects in Groups 1 5 will complete the Use the Product Again questionnaire at 21:30 (± 30 minutes) on Day 7. Subjects in Group 1 will complete Use the Product Again questionnaire for cigarettes. Subjects in Groups 2 and 3 will complete both Use the Product Again questionnaire for cigarettes and VERVE® products. Subjects

in Groups 4 and 5 will complete Use the Product Again questionnaire for VERVE® products.

## 7.1.4.2 Analysis Variables

## **QSU-Brief**

According to the literature<sup>1</sup>, the factor scores for the QSU-Brief will be calculated as follows.

- Factor 1 (anticipation of pleasure from smoking): average of items 1, 3, 6, 7, and 10.
- Factor 2 (relief of nicotine withdrawal): average of items 2, 4, 5, 8, and 9.

The following variable will be determined for each factor score.

• Change from pre-product use score  $(07:00 \pm 30 \text{ min})$  to post-product use score  $(21:30 \pm 30 \text{ min})$ , i.e. post-product use score minus pre-product use score, on each day

### Modified Cigarette Evaluation Questionnaires

Responses on the 7-point scales for each mCEQ (mCEQ-V for days in which VERVE® products are used and mCEQ-C for days in which subject's OB cigarettes are used) will be treated as continuous variables and the following factor scores will be calculated according to the literature<sup>2</sup>:

- Smoking satisfaction: average of the response scores from questions 1, 2, and 12;
- Psychological reward: average of the response scores from questions 4 to 8;
- Aversion: average of the response scores from questions 9 and 10;
- Enjoyment of sensation: response score from question 3;
- Craving Reduction: response score from question 11.

The following variable will be determined for each factor score.

Actual score

### Use Product Again Questionnaires

The analysis variable will be the response VAS score to the Use the Product Again questionnaire for each product. In addition, responses to Use the Product Again questionnaire will also be treated as bipolar variable and used as an analysis variable. The bipolar score is calculated by subtracting 50 from the original VAS score, then categorizing into three categories: -50 to <0, 0, and >0 to 50.

## 7.2 Data Summary and Presentation

The descriptive statistics tables for blood and urine biomarkers, products used per day, and subjective effects will be generated with the following level of precision for the summary statistics:

The derived values (amount excreted in urine biomarkers, change and percent change from baseline) will have two decimal points.

- Number of observations (n)/number of missing values (n missing) without a decimal:
- Mean/median with one more decimal/significant figure than minimum/ maximum;
- Q1 and Q3 with one more decimal/significant figure than minimum/ maximum;
- Standard deviation/standard error of the mean (SD/SEM) with one more decimal/significant figure than mean/median.
- Coefficient of variation (CV%) with one decimal;
- Minimum/maximum in same precision as in the database
- 95% confidence intervals (CI) with one more decimal/significant figure than minimum/ maximum

## 7.2.1 Demographic Summary

Descriptive statistics will be summarized for continuous demographics variables (e.g., age, weight, height, and BMI) and frequency counts will be tabulated for categorical demographics variables (e.g., gender, ethnicity, race, income level, and highest education grade level) by study group, and overall. The variable BMI is calculated from the weight and height collected at the Screening assessment and age is calculated from the date of the Screening visit. Subjects only enrolled in the product trial period (dropped prior to randomization) will be summarized separately as a group.

The Safety, mITT and PP populations will be used for this summary.

### 7.2.2 Smoking History

CPD including Days -2 through -1 collected on site, years of smoking (calculated from Screening date), Fagerström Test for Cigarette Dependence scores (individual questions and total score), and usual brand, brand style, flavor, and cigarette size reported at Screening will be listed. Descriptive statistics will be summarized by study group and overall for continuous variables and frequency counts and percentage will be presented for categorical variables. Subjects only enrolled in the product trial period will be summarized separately as a group.

The Safety, mITT and PP populations will be used for this summary.

#### 7.2.3 Urine BOE

Urine biomarker concentration (including each component of NE), urine creatinine concentration, and the creatinine-adjusted urine biomarker concentration will be listed by subject and study day for all urine biomarkers. All BLQ values will be presented as "BLQ" in the listings.

Urine biomarker mass excreted per 24 hours, absolute change from baseline and percent change from baseline of total mass excreted per 24 hours, and creatinine-adjusted urine biomarker concentrations, will be summarized by group and study day for all urine biomarkers using descriptive statistics (n, n missing, mean, SD, CV%, SEM, minimum, median, maximum, and 95% CI). The descriptive statistics will be provided for both mITT and PP populations.

### 7.2.4 Blood BOE

Blood biomarker concentrations will be listed by subject and study visit for COHb. All BLQ values for COHb will be presented as "BLQ" in the listings.

Blood biomarker concentration, absolute change from baseline blood biomarker concentration, and percent change from baseline biomarker concentration will be summarized by group and study day using descriptive statistics (n, n missing, mean, SD, CV%, SEM, minimum, median, maximum, and 95% CI). BLOQ COHb saturation will be treated as one-half the LLOQ. The descriptive statistics will be provided for both mITT and PP populations.

#### 7.2.5 Product Use

#### Product Use

Number of CPD smoked per day (Groups 1, 2, and 3, only), number of VPD per day (Groups 2, 3, 4, and 5 only), average duration of VERVE® product used per use each day (Groups 2, 3, 4, and 5 only), and total duration of VERVE® product use per Day (Groups 2, 3, 4, and 5 only) will be listed by subject and study day and summarized by group and study day using descriptive statistics (n, n missing, mean, SD, CV%, SEM, minimum, Q1, median, Q3, maximum and 95% CI). The start time of VERVE producct use along time of the day (x-axis, 7:00 to 23:00) by group (y-axis, Group 2, 3, 4, 5) for Day 1, 5, 7 (one plot per day) will be plotted.

Product use analyses will be performed on the mITT dataset.

## 7.2.6 Questionnaires

The responses and the factor scores from the QSU-Brief will be listed by subject, study day and collection time. Factor scores (original scores, and change from pre-use scores) will be summarized by group, day and collection time using descriptive statistics (n, n missing, mean, SD, CV%, SEM, minimum, Q1, median, Q3, maximum, and 95% CI).

The mCEQ will be considered as a 7-point scale and treated as a continuous variable. The responses from mCEQ-C or mCEQ-V and factor scores will be listed by subject and study day. The factor scores will be summarized by group and study day using descriptive statistics (n, n missing, mean, SD, CV%, SEM, minimum, Q1, median, Q3, maximum and 95% CI).

Responses to Use the Product Again questionnaire recorded as VAS scores will be treated as bipolar variable and summarized by study group, study product and category using frequency count tables. The original response VAS score and bipolar score for the Use the Product Again questionnaire will be summarized using descriptive statistics (n, n missing, mean, SD, CV%, SEM, minimum, Q1, median, Q3, maximum and 95% CI).

These analyses will be performed on the mITT dataset.

# 7.3 Statistical Analyses

## 7.3.1 Primary Endpoint Analysis

A linear mixed model for repeated measures (MMRM) analysis will be used for comparing each test group (Groups 2-5) to the control group (Group 1 and Group 6) in the primary endpoint (24-hour total urinary NNAL (mg/24 hours) excreted on Day 7). In the model, study group, study day, and study group by study day interaction, and gender are the fixed effect factors. The baseline value of the response biomarker is the covariate. A restricted maximum likelihood estimation method will be applied and several covariance structures will be tried. Five candidate covariance structures will be considered: compound symmetry, 1st order autoregressive, 1st order autoregressive with a random subject effect, unstructured and Toeplitz. The most appropriate covariance structure will be determined based on the AIC criteria (the covariance structure with the smallest AIC will be chosen). The least-square mean, 95% confidence interval and p-value will be provided for the study groups. The leastsquare mean difference, 95% confidence interval and p-value will be provided for the study group comparisons. Pairwise comparisons (Group 2 vs. Group 1, Group 3 vs. Group 1, Group 4 vs. Group 1, Group 5 vs. Group 1, Group 2 vs. Group 6, Group 3 vs. Group 6, Group 4 vs. Group 6, and Group 5 vs. Group 6,) will be performed using a Dunnett's test at a 2-sided significance level of 0.05 to adjust for multiplicity. Group 1 & 6 will be considered as the control groups. The test is for each of the other groups to compare with the control groups. The analysis will be conducted on the mITT and PP datasets.

The following SAS codes will be used to perform the analysis.

```
Proc mixed data=<>;
Class subject gender group day;
Model response = gender group day group*day baseline/ddfm=kr;
Repeated day/type=<type> subject=subject;
LSmeans group*day/CL alpha=0.05 pdiff dunnett ('1'*Day 7, '6'*Day 7);
```

Run;

Note: This model will include both the Day 7 value (primary endpoint) and interim time points (Day 5, secondary endpoint). The above analysis will also output the residual diagnosis to check for normality and to identify outliers).

## 7.3.1.1 Multiplicity adjustment

There is one primary analysis variable. No multiplicity adjustment will be done among biomarkers. For the test groups compared to the reference groups for each biomarker, Dunnett's method will be used for the adjustment of multiple comparisons.

# 7.3.1.2 Dealing with non-normality

A standard residual analysis using Proc Mixed procedure will be used to examine validity of normality assumptions for the primary endpoint. A natural logarithmic transformation might be applied to the endpoint in the linear mixed model with repeated measurements if the normality assumption does not hold. Square Root transformation will be used for urine mutagenicity statistical analysis.

## 7.3.2 Secondary Endpoint Analysis

The same statistical analysis model defined in the primary analysis Section 7.3.1 will also be used to make same comparisons as the primary endpoint (i.e. total NNAL on Day 7) for the secondary biomarker endpoints listed in Section 2.4.

These analyses will be conducted on the mITT and PP datasets.

## 7.3.3 Subjective Effects

Similar statistical comparison analysis (defined in 7.3.1) will be preformed on QSU-brief change from pre-use score and mCEQ original scores (mCEQ-C, among Group 1, 2, and 3; mCEQ-V, among Groups 2, 3, 4, and 5). The comparisons interested for QSU-brief will be the test groups (Groups 2-5) versus the continue smoking group (Group 1) and test groups (Groups 2-5) versus the tobacco cessation Group. The comparisons interested for mCEQ-C will be the dual use groups (Groups 2-3) versus the continue smoking group (Group 1). The comparisons interested for mCEQ-V will be the dual use groups (Groups 2-3) versus the exclusive use group (Groups 4 -5) [i.e. Group 2 vs Group 4 and Group 3 vs Group 5].

This analysis will be conducted on the mITT datasets. No multiple adjustment will be performed for subject effect scores.

## 7.3.4 Sensitivity Analysis

## 7.3.4.1 Analysis Variables for Sensitivity Analysis

The sensitivity analysis will be performed for primary endpoint (24-hour total urinary NNAL (ng/24 hours) excreted on Day 7).

## 7.3.4.2 Handling of Missing Data

Two methods (last observation carried forward and multiple imputation) will be tested for the handling of missing data for the primary endpoint if the percentage of missing data is larger than 5% in the mITT population. For all other analyses, data will not be imputed. Baseline is not expected to be missing for the mITT population.

Multiple imputation will be conducted to impute the missing data values for the primary endpoints (24-hour total urinary NNAL (ng/24 hours) excreted on Day 7). The imputation starts with using SAS procedure Proc MI to generate (n=m) completed data sets. Then each data set will be analyzed with SAS procedure Proc Mixed to generate m point estimates and standard errors for the model parameters. Finally, SAS procedure Proc Mianlyze will be used to combine the estimation results

The Following SAS codes will be used for imputation and analysis.

1) use PROC MI to impute the missing data;

```
proc mi data=... seed=... nimpute=200 out=miout noprint; mcmc; var biomarker_baseline biomarker_Day5 biomarker_Day7; run;
```

2) use PROC MIXED to model the multiple imputed datasets:

```
proc mixed data=miout order=internal; where day=7; by _imputation_; class subject gender group; model biomarker = gender group baseline/ddfm=kr; lsmeans group / alpha=0.05 CL pdiff; ods output lsmeans=lsmnout; ods output diffs=diff; run;
```

3) use PROC MIANALYZE to generate the int (lsmnoutmi, diffmi) from the multiple estimates (lsmnout, diff).

```
proc sort data=lsmnout;by group _imputation_;run; proc mianalyze data=lsmnout alpha=0.05;
```

```
by group;
modeleffects group;
ods output ParameterEstimates=lsmnoutmi;
stderr stderr;
run;

proc sort data=diff;by group _imputation_;run;
proc mianalyze data=diff alpha=0.05;
by group;
modeleffects group;
ods output ParameterEstimates=diffmi;
stderr stderr;
run;
```

# 7.3.4.3 Examining Influence of Outliers

Data outliers will be examined through Proc Mixed model residual diagnosis (+/- 4 studentized residuals). The outlier test results will be conducted for the primary endpoint (24-hour total urinary NNAL (ng/24 hours) excreted on Day 7). A sensitivity analysis by excluding outliers will be performed for the primary analysis variable if any outliers are found using the above criteria.

## 7.3.4.4 Handling BLQ values

Values below the limit of quantitation (BLQ) for nicotine and its metabolites, COHb, and other urine biomarkers will be presented in the data listings as BLQ. Values BLQ for nicotine and metabolites will be set to one-half of the limit of quantitation prior to use in the calculation of nicotine equivalents and data analysis of NE. Values BLQ for other urine biomarkers and COHb will be set to one-half of the LLOQ prior to data analysis. A sensitivity analysis of the primary endpoint (24-hour total urinary NNAL (ng/24 hours) excreted on Day 7) analysis will be conducted by setting the BLQ value to the LLOQ if the percentage of values that are BLQ is greater than 5% of observations.

Approximate LLOQ values for each analyte are shown in the table below. LLOQs will be reported out to the most current validation data and included in the bioanalytical report.

| Analyte | LLOQ |
|--------------------------------------|------------|
| Nicotine | 50.0 ng/mL |
| Cotinine | 50.0 ng/mL |
| trans-3'-hydroxycotinine | 50.0 ng/mL |
| nicotine glucuronide | 50.0 ng/mL |
| cotinine glucuronide | 200 ng/mL |
| trans-3'-hydroxycotinine glucuronide | 200 ng/mL |

| NNN | 0.500 pg/mL |
|------------|-------------|
| NNAL | 2.00 pg/mL |
| 2-AN | 1.7 pg/mL |
| HEMA | 0.2 ng/mL |
| 3-HMPMA | 5 ng/mL |
| 3-HPMA | 25 ng/mL |
| CEMA | 0.25 ng/mL |
| 4-ABP | 1.5 pg/mL |
| S-PMA | 0.02 ng/mL |
| 2-HPMA | 2.5 ng/mL |
| AAMA | 10 ng/mL |
| GAMA | 1 ng/mL |
| 2-MHBMA | 0.129 ng/mL |
| 2-OHFle | 0.05 ng/mL |
| 2-Naphthol | 0.10 ng/mL |
| 1-OHP | 0.01 ng/mL |
| Creatinine | 30 μg/mL |
| СОНЬ | 0.2% |

### 8. SAFETY

No inferential statistics will be performed on the safety data.

All clinical safety data will be listed by subject. Continuous variables will be summarized using n, mean, SD, median, minimum, and maximum. Frequency counts will be reported for all categorical data.

Decimal point will be presented as follows:

- n will be presented without decimal;
- Minimum/maximum in same precision as in the database;
- Mean/median in one more decimal than minimum/maximum;
- SD in one more decimal than mean/median.

Where individual data points are missing because of dropouts or other reasons, the data will be summarized based on reduced denominators.

## 8.1 Subject Disposition

The number of subjects enrolled, the number who completed the study, and the number who did not complete the study (overall and reasons for early withdrawal) will be tabulated by study group and overall. A listing of subjects who discontinued the study prematurely will also be presented. Screen failure subjects and subjects only enrolled in the product trial period will be summarized separately.

#### 8.2 Adverse Events

Adverse events will be coded (to the lowest level term) with the Medical Dictionary for Regulatory Activities (MedDRA®) version 20.0.

A study product use-emergent AE is defined as an AE that is starting or worsening at the time of or after study product administration.

All events captured in the database will be listed in by-subject data listings. However, only study product use-emergent adverse events will be summarized.

Frequencies of subjects with study product use-emergent AEs, regardless of relationship to study product will be summarized by study group and sorted by system organ class. Frequencies of subjects with study product use-emergent serious adverse events will be likewise summarized. Frequencies of study product use-emergent adverse events will be summarized by severity and relationship to study product. Adverse events occurred during the product trial period will be summarized separately as a group.

## 8.3 Clinical Laboratory

Clinical laboratory evaluations (clinical chemistry, hematology, and urinalysis) will be performed at Screening and at End-of-Study or Early Termination.

Descriptive statistics will be reported for numeric clinical data by study group and time point. Rechecked values prior to randomization will be used in calculating summary statistics. Normal ranges will be listed by site. Subjects only enrolled in the product trial period will be summarized separately.

Out of normal range and clinically significant laboratory values will be listed by subject.

A urine cotinine test will be completed at Screening. Urine drug tests and alcohol breath tests will be completed at Screening. Serum pregnancy tests will be completed at Screening and urine pregnancy tests will be completed at Check-in. Results for these tests will be listed as "Negative" or "Positive."

## 8.4 Vital Signs

Vital signs (respiration rate, pulse rate, blood pressure, and oral temperature) will be measured at screening, at Check-in, and at the End-of-Study or upon Early Termination.

Descriptive statistics will be reported for vital sign measurements (blood pressure, pulse, respiration, and temperature) by study group and time point. Post randomization rechecks will not be used for calculation of descriptive statistics. Subjects only enrolled in the product trial period will be summarized separately.

#### 8.5 ECG

A 12-lead ECG will be obtained during screening and listed by subject.

#### **8.6** Concomitant Medications

All concomitant medications recorded during the study will be coded using the WHO Drug Dictionary (WHODD) version 01MAR2018 and listed by subject.

## 8.7 Physical Examination

Physical examinations will be performed at Screening. A brief physical examination (symptom driven) may be performed at Check-in and End of Study (or Early Termination). Physical examinations will be listed by subject and time point of collection. Changes in physical examinations (if any) will be described in the text of the final report.

### 9. SUMMARY OF CHANGES FROM PROTOCOL-PLANNED ANALYSIS

The analyses described in this SAP are aligned with those analyses described in the protocol with the following changes for statistical analysis.

- 1. Mixed model with repeated measurement instead of mixed model will be used in the analysis for biomarker statistical analysis as there are two response values (Days 5 and 7) for each subject.
- 2. Emax for Use Product Again questionnaire was mentioned in the protocol. As the Use Product Again questionnaire will only be conducted at Day 7 and only one response value for each subject, no maximum value will be available. The analysis will be performed based on the original response.
- 3. The statistical analysis model for Use Product Again questionnaire was modified based on the study design and data collection.

## 10. SUMMARY TABLES AND FIGURES

Summary tables and figures are numbered following the International Conference on Harmonization (ICH) structure. Please note that all summary tables and figures will be generated using SAS® Version 9.3 or higher.

The following is a list of table numbers and titles that will be included as summary tables:

## 14.1 Demographic Data Summary Tables

Table 14.1.1.1 Summary of Disposition by Study Group and Overall

Table 14.1.1.2 Summary of Disposition for Screen Failures

- Table 14.1.2 Demographic Summary by Study Group and Overall Table 14.1.3 Smoking History by Study Group and Overall
- 14.2 Data Summary Tables and Figures for Biomarkers, Product Use, and Questionnaire Reponses

## 14.2.1 Urine and Blood Biomarkers Tables

| Primary and Secondary Biomarker endpoints | |
|---|---|
| Total Urine NNAL | |
| Table 14.2.1.1.1.1 | Summary of Total Urine NNAL 24-Hour Excreted (ng/24 hour) by Study Group and Study Day (mITT Population) |
| Table 14.2.1.1.1.2 | Summary of Total Urine NNAL 24-Hour Excreted (ng/24 hour) by Study Group and Study Day (PP Population) |
| Table 14.2.1.1.2.1 | Summary of Total Urine NNAL 24-Hour Excreted Absolute Change From Baseline (ng/24 hour) by Study Group and Study Day (mITT Population) |
| Table 14.2.1.1.2.2 | Summary of Total Urine NNAL 24-Hour Excreted Absolute Change From Baseline (ng/24 hour) by Study Group and Study Day (PP Population) |
| Table 14.2.1.1.3.1 | Summary of Total Urine NNAL 24-Hour Excreted Percent Change From Baseline (%) by Study Group and Study Day (mITT Population) |
| Table 14.2.1.1.3.2 | Summary of Total Urine NNAL 24-Hour Excreted Percent Change From Baseline (%) by Study Group and Study Day (PP Population) |
| Table 14.2.1.1.4.1 | Summary of Total Urine NNAL Adjusted for Urine Creatinine (ng/g creatinine) by Study Group and Study Day (mITT Population) |
| Table 14.2.1.1.4.2 | Summary of Total Urine NNAL Adjusted for Urine Creatinine (ng/g creatinine) by Study Group and Study Day (PP Population) |
| Table 14.2.1.1.5.1 | Statistical Summary of Total Urine NNAL 24-Hour Excreted (ng/24 hour) by Study Group and Study Day (mITT Population) |

Day (mITT Population)

Statistical Comparisons of Total Urine NNAL 24-Hour

Excreted (ng/24 hour) Between Study Groups by Study

Table 14.2.1.1.5.2

| rioject CA24303 | |
|---|---|
| Table 14.2.1.1.6.1 | Statistical Summary of Total Urine NNAL 24-Hour Excreted (ng/24 hour) by Study Group and Study Day (PP Population) |
| Table 14.2.1.1.6.2 | Statistical Comparisons of Total Urine NNAL 24-Hour Excreted (ng/24 hour) Between Study Groups by Study Day (PP Population) |
| Table 14.2.1.1.7.1 | Statistical Summary of Total Urine NNAL 24-Hour Excreted (ng/24 hour) by Study Group (mITT Population with Imputation of Missing Data Using Last Observation Carried Forward Method) (Note: This analysis will only be performed if the percentage of missing values is greater than 5% of observations.) |
| Table 14.2.1.1.7.2 | Statistical Comparisons of Total Urine NNAL 24-Hour Excreted (ng/24 hour) Study Groups (mITT Population with Imputation of Missing Data Using Last Observation Carried Forward Method) (Note: This analysis will only be performed if the percentage of missing values is greater than 5% of observations.) |
| Table 14.2.1.1.8.1 | Statistical Summary of Total Urine NNAL 24-Hour Excreted (ng/24 hour) by Study Group (mITT Population with Imputation of Missing Data Using Multiple Imputation by SAS MI Procedure) (Note: This analysis will only be performed if the percentage of missing values is greater than 5% of observations.) |
| Table 14.2.1.1.8.2 | Statistical Comparisons of Total Urine NNAL 24-Hour Excreted (ng/24 hour) Between Study Groups (mITT Population with Imputation of Missing Data Using Multiple Imputation by SAS MI Procedure) (Note: This analysis will only be performed if the percentage of missing values is greater than 5% of observations.) |
| Table 14.2.1.1.9.1 | Summary of Total Urine NNAL 24-Hour Excreted (ng/24 hour) by Study Group and Study Day (mITT Population with Outliers Excluded) |
| Table 14.2.1.1.9.2 | Statistical Summary of Total Urine NNAL 24-Hour Excreted (ng/24 hour) at Day 7 by Study Group (mITT Population with Outliers Excluded) |
| Table 14.2.1.1.9.3 | Statistical Comparisons of Total Urine NNAL 24-Hour Excreted (ng/24 hour) at Day 7 Between Study Groups (mITT Population with Outliers Excluded) |

Table 14.2.1.1.10.1 Statistical Summary of Total Urine NNAL 24-Hour

Excreted (ng/24 hour) at Day 7 by Study Group (mITT

Population with BLQ values set to the LLOQ) (Note: This analysis will only be performed if the percentage of values that are BLQ is greater than 5% of observations.)

Table 14.2.1.1.10.2 Statistical Comparisons of Total Urine NNAL 24-Hour Excreted (ng/24 hour) at Day 7 Between Study Groups (mITT Population with BLQ values set to the LLOQ) (Note: This analysis will only be performed if the percentage of values that are BLQ is greater than 5% of observations.)

For the following urine biomarkers, tables similar to those for Total Urine NNAL will be created as appropriate and numbered as specified:

#### **Urine NNN Tables**

Tables 14.2.1.2.1.1 through 14.2.1.2.6.2

## Urine Nicotine Equivalents Tables

Tables 14.2.1.3.1.1 through 14.2.1.3.6.2

### **Urine 2-AN Tables**

Tables 14.2.1.4.1.1 through 14.2.1.4.6.2

#### Urine 4-ABP Tables

Tables 14.2.1.5.1.1 through 14.2.1.5.6.2

#### Urine HEMA Tables

Tables 14.2.1.6.1.1 through 14.2.1.6.6.2

### Urine CEMA Tables

Tables 14.2.1.7.1.1 through 14.2.1.7.6.2

### **Urine S-PMA Tables**

Tables 14.2.1.8.1.1 through 14.2.1.8.6.2

#### **Urine 3-HMPMA Tables**

Tables 14.2.1.9.1.1 through 14.2.1.9.6.2

## Urine 3-HPMA Tables

Tables 14.2.1.10.1.1 through 14.2.1.10.6.2

### Urine 2-HPMA Tables

Tables 14.2.1.11.1.1 through 14.2.1.11.6.2

#### Urine AAMA Tables

Tables 14.2.1.12.1.1 through 14.2.1.12.6.2

#### Urine GAMA Tables

Tables 14.2.1.13.1.1 through 14.2.1.13.6.2

## **Urine 2-MHBMA Tables**

Tables 14.2.1.14.1.1 through 14.2.1.14.6.2

## **Urine 2-OHFle Tables**

Tables 14.2.1.15.1.1 through 14.2.1.15.6.2

## Urine 2-Naphthol Tables

Tables 14.2.1.16.1.1 through 14.2.1.16.6.2

### **Urine 1-OHPhe Tables**

Tables 14.2.1.17.1.1 through 14.2.1.17.6.2

### **Urine 1-OHP Tables**

Tables 14.2.1.18.1.1 through 14.2.1.18.6.2

## Urine Mutagenicity Tables

Tables 14.2.1.19.1.1 through 14.2.1.19.6.2

### **Blood COHb Tables**

| Table 14.2.1.20.1.1 | Summary | of Blood | COHb | (% | Saturation) | by | Study |
|---|---|---|---|---|---|---|---|
| | Group and | Study Day | (mITT | Pop | ulation) | | |

- Table 14.2.1.20.1.2 Summary of Blood COHb (% Saturation) by Study Group and Study Day (PP Population)
- Table 14.2.1.20.2.1 Summary of Blood COHb Absolute Change From Baseline (% Saturation) by Study Group and Study Day (mITT Population)
- Table 14.2.1.20.2.2 Summary of Blood COHb Absolute Change From Baseline (% Saturation) by Study Group and Study Day (PP Population)

| Table 14.2.1.20.3 | 3.1 Summary of Blood COHb Percent Change From Baseline (%) by Study Group and Study Day (mITT Population) |
|---|---|
| Table 14.2.1.20.3 | 3.2 Summary of Blood COHb Percent Change From Baseline (%) by Study Group and Study Day (PP Population) |
| Table 14.2.1.20.4 | 4.1 Statistical Summary of Blood COHb (% Saturation) by Study Group and Study Day (mITT Population) |
| Table 14.2.1.20.4 | 4.2 Statistical Comparisons of Blood COHb (% Saturation) Between Study Groups by Study Day (mITT Population) |
| Table 14.2.1.20.5 | 5.1 Statistical Summary of Blood COHb (% Saturation) by Study Group and Study Day (PP Population) |
| Table 14.2.1.20.5 | |
| 14.2.2 Product | Use |
| Table 14.2.2.1 | Summary of Number of Cigarettes Smoked Per Day by Study Group and Study Day (mITT Population) |
| Table 14.2.2.2 | Summary of VERVE Product Used Per Day by Stud<br>Group and Study Day (mITT Population) |
| Table 14.2.2.3 | Summary of Average Duration of VERVE Product Used<br>Per Use by Study Group and Study Day (mITT<br>Population) |
| Table 14.2.2.4 | Summary of Total Duration of VERVE Product Per Day by Study Group and Study Day (mITT Population) |
| 14.2.3 Subjective Effective | et Questionnaires |
| QSU-Brief Ques | tionnaire |
| Table 14.2.3.1.1 | Summary of QSU-Brief Factor Scores and Change from<br>Pre Product Use by Study Group and Study Day (mITT<br>Population) |
| Table 14.2.3.1.2. | Statistical Summary of QSU-Brief Factor Change from Pre Product Use Scores by Study Group and Study Day (mITT Population) |
| Table 14.2.3.1.2. | 2 Statistical Comparisons of QSU-Brief Factor Change<br>from Pre Product Use Scores Between Study Groups by<br>Study Day (mITT Population) |
| mCEQ | - · · · |
| Table 14.2.3.2.1 | Summary of mCEQ Factor Scores by Study Group and |

Study Day (mITT Population)

| Table 14.2.3.2.2.1 | Statistical Summary of mCEQ-C Factor Scores by Study<br>Group and Study Day (mITT Population) |
|---|---|
| Table 14.2.3.2.2.2 | Statistical Comparisons of mCEQ-C Factor Scores<br>Between Study Groups by Study Day (mITT Population) |
| Table 14.2.3.2.3.1 | Statistical Summary of mCEQ-V Factor Scores by Study<br>Group and Study Day (mITT Population) |
| Table 14.2.3.2.3.2 | Statistical Comparisons of mCEQ-V Factor Scores<br>Between Study Groups by Study Day (mITT Population) |

## Use Product Again

- Table 14.2.3.3.1 Frequency of Response to Use the Product Again VAS Scores by Study Group and Study Product (mITT Population)
- Table 14.2.3.3.2 Summary of Response to Use the Product Again VAS Scores by Study Group and Study Product (mITT Population)
- Table 14.2.3.3.3 Summary of Response to Use the Product Again Bipolar Scores by Category, Study Group and Study Product (mITT Population)

## 14.2.4 Biomarker Figures (mITT, PP Populations)

| Total Urine NNAL Count Figures | |
|---|---|
| Figure 14.2.4.1.1 | Box Plot of Total Urine NNAL 24-Hour Excreted (ng/24 hour) at Baseline and Day 7 by Study Group (mITT Population) |
| Figure 14.2.4.1.2 | Box Plot of Total Urine NNAL 24-Hour Excreted (ng/24 hour) at Baseline and Day 7 by Study Group (PP Population) |
| Figure 14.2.4.1.3 | Box Plot of Total Urine NNAL 24-Hour Excreted (ng/24 hour) at Baseline and Day 5 by Study Group (mITT Population) |

For the following urine biomarkers, figuress similar to those for Total Urine NNAL will be created as appropriate and numbered as specified:

## **Urine NNN Figures**

Figures 14.2.4.2.1 through 14.2.4.2.3

## Urine Nicotine Equivalents Figures

Figures 14.2.4.3.1 through 14.2.4.3.3

### **Urine 2-AN Figures**

Figures 14.2.4.4.1 through 14.2.4.4.3

## Urine 4-ABP Figures

Figures 14.2.4.5.1 through 14.2.4.5.3

## Urine HEMA Figures

Figures 14.2.4.6.1 through 14.2.4.6.3

## Urine CEMA Figures

Figures 14.2.4.7.1 through 14.2.4.7.3

### **Urine S-PMA Figures**

Figures 14.2.4.8.1 through 14.2.4.8.3

## Urine 3-HMPMA Figures

Figures 14.2.4.9.1 through 14.2.4.9.3

## Urine 3-HPMA Figures

Figures 14.2.4.10.1 through 14.2.4.10.3

### *Urine 2-HPMA Figures*

Figures 14.2.4.11.1 through 14.2.4.11.3

## Urine AAMA Figures

Figures 14.2.4.12.1 through 14.2.4.12.3

## Urine GAMA Figures

Figures 14.2.4.13.1 through 14.2.4.13.3

## Urine 2-MHBMA Figures

Figures 14.2.4.14.1 through 14.2.4.14.3

## *Urine 2-OHFle Figures*

Figures 14.2.4.15.1 through 14.2.4.15.3

## Urine 2-Naphthol Figures

Figures 14.2.4.16.1 through 14.2.4.16.3
## Urine 1-OHPhe Figures

Figures 14.2.4.17.1 through 14.2.4.17.3

#### **Urine 1-OHP Figures**

Figures 14.2.4.18.1 through 14.2.4.18.3

# Urine Mutagenicity Figures

Figures 14.2.4.19.1 through 14.2.4.19.3

#### Whole Blood COHb Figures

| Figure 14.2.4.20.1 | Box Plot of Whole Blood COHb (% Saturation) at |
|--------------------|-----------------------------------------------------|
| | Baseline and Day 7 by Study Group (mITT Population) |
| Figure 14.2.4.20.2 | Box Plot of Whole Blood COHb (% Saturation) at |
| | Baseline and Day 7 by Study Group (PP Population) |
| Figure 14.2.4.20.3 | Box Plot of Whole Blood COHb (% Saturation) at |
| | Baseline and Day 5 by Study Group (mITT Population) |

# **14.2.5 Product Use Figures (mITT Populations)**

| Figure 14.2.5.1 | Start Time of VERVE Product Use Along Time of the |
|---|---|
| | Day by Study Group (Day 1) (mITT Population) |
| Figure 14.2.5.2 | Start Time of VERVE Product Use Along Time of the Day by Study Group (Day 5) (mITT Population) |
| Figure 14.2.5.3 | Start Time of VERVE Product Use Along Time of the Day by Study Group (Day 7) (mITT Population) (mITT Population) |

Note: The x-axis will be the time of the day (from 7:00 to 23:00), the y-axis will have 4 ticks for the 4 groups (Groups 2-5). All the start times from all the subjects in the same group will form a single horizontal dotted line. The dotted line will be dense at certain timepoints when the subjects are using the VERVE product at the same time, otherwise the dotted line is loose.

## 14.3 Safety Data Summary Tables

# 14.3.1 Displays of Adverse Events

- Table 14.3.1.1 Adverse Event Frequency by Study Group Number of Subjects Reporting the Event (% of Subjects Who Received Study Product or in Study Group)
- Table 14.3.1.2 Adverse Event Frequency by Study Group Number of Adverse Events (% of Total Adverse Events)
- Table 14.3.1.3 Adverse Event Frequency by Study Group, Severity, and Relationship to Study Product Number of Subjects Reporting Events
- Table 14.3.1.4 Adverse Event Frequency by Study Group, Severity, and Relationship to Study Product Number of Adverse Events

# 14.3.2 Listings of Deaths, other Serious and Significant Adverse Events

Table 14.3.2.1 Serious Adverse Events (if no serious adverse event occurred, a statement 'No serious adverse event is reported' will be in the table)

# 14.3.3. Narratives of Deaths, other Serious and Certain other Significant Adverse Events

### 14.3.4. Abnormal Laboratory Value Listing (each subject)

- Table 14.3.4.1 Out-of-Range Values and Recheck Results Serum Chemistry
- Table 14.3.4.2 Out-of-Range Values and Recheck Results Hematology
- Table 14.3.4.3 Out-of-Range Values and Recheck Results Urinalysis

# 14.3.5. Displays of Other Laboratory, Vital Signs, Electrocardiogram, Physical Examination, and Other Safety Data

- Table 14.3.5.1 Clinical Laboratory Summary Serum Chemistry
- Table 14.3.5.2 Clinical Laboratory Summary Hematology
- Table 14.3.5.3 Clinical Laboratory Summary Urinalysis
- Table 14.3.5.4 Vital Sign Summary

#### 11. DATA LISTING TITLES AND NUMBERS

Note: Hepatitis and HIV results that are provided by the clinical laboratory will not be presented in subject data listings and will not be included in any database transfer.

Data listings are numbered following the ICH structure. The following is a list of appendix numbers and titles that will be included as data listings:

#### 16.1. Study Information

Appendix 16.1.10.1 Clinical Laboratory Reference Ranges

## 16.2. Subject Data Listings

#### 16.2.1. Subject Discontinuation

Appendix 16.2.1.1 Subject Disposition and Discontinuation (Randomized)

Appendix 16.2.1.2 Subject Disposition and Discontinuation (Product Trial)

Appendix 16.2.1.3 Subject Disposition and Discontinuation (Screen Failures)

Appendix 16.2.1.4 Subject Population information

#### 16.2.2. Protocol Deviations

Appendix 16.2.2 Protocol Deviations

# 16.2.3. Subjects Excluded from Biomarker Analysis

Appendix 16.2.3 Subjects Excluded from Biomarker Analysis

Note: Appendices 16.2.2 and 16.2.3 are generated in Microsoft® Word® for inclusion in the CSR.

## 16.2.4. Demographic Data

| Appendix 16.2.4.1.1 | Demographics (I of II) |
|---------------------|-------------------------------------------------|
| Appendix 16.2.4.1.2 | Demographics (II of II) |
| Appendix 16.2.4.1.3 | Subject Characteristics |
| Appendix 16.2.4.2.1 | Physical Examination (I of II) |
| Appendix 16.2.4.2.2 | Physical Examination (II of II) |
| Appendix 16.2.4.2.3 | Physical Examination Descriptions |
| Appendix 16.2.4.3 | Medical History |
| Appendix 16.2.4.4.1 | Tobacco/Nicotine Product Use History (I of II) |
| Appendix 16.2.4.4.2 | Tobacco/Nicotine Product Use History (II of II) |
| Appendix 16.2.4.5 | Fagerstrom Test for Cigarette Depedence |

# 16.2.5. Compliance Data

| Appendix 16.2.5.1 | Inclusion / | Exclusion | Criteria | Not Met |
|-------------------|-------------|-----------|----------|---------|
|-------------------|-------------|-----------|----------|---------|

Appendix 16.2.5.2.1 Product Trial

Appendix 16.2.5.2.2 In-Clinic Product Use

Appendix 16.2.5.2.3 Max CPD

Appendix 16.2.5.3.1 24-Hour Urine Collection

Appendix 16.2.5.3.2 Urine Samples

| Appendix | 16.2.5.4 | Carboxyhemoglobin Blood Collection |
|---|---|---|
| Appendix | 16.2.5.5 | Prior and On-Study Concomitant Medications |
| 16.2.6. | Individual | Response Data |
| Appendix | 16.2.6.1 | Total Urine NNAL |
| Appendix | | Urine NNN |
| Appendix | | Urine Nicotine and Metabolites Concentrations |
| Appendix | | Urine Nicotine Equivalents |
| Appendix | | Urine 2-AN |
| Appendix | 16.2.6.5 | Urine 4-ABP |
| Appendix | | Urine HEMA |
| Appendix | | Urine CEMA |
| Appendix | | Urine S-PMA |
| Appendix | | Urine 3-HMPMA |
| Appendix | 16.2.6.10 | Urine 3-HPMA |
| Appendix | 16.2.6.11 | Urine 2-HPMA |
| Appendix | 16.2.6.12 | Urine AAMA |
| Appendix | 16.2.6.13 | Urine GAMA |
| Appendix | 16.2.6.14 | Urine 2-MHBMA |
| Appendix | 16.2.6.15 | 2-OHFle |
| Appendix | 16.2.6.16 | Urine 2-Naphthol |
| Appendix | 16.2.6.17 | Urine 1-OHPhe |
| Appendix | 16.2.6.18 | Urine 1-OHP |
| Appendix | 16.2.6.19 | Whole Blood COHb |
| Appendix | 16.2.6.20.1 | Cigarettes Used per Day |
| Appendix | 16.2.6.20.2 | VERVE Product Used per Day |
| Appendix | 16.2.6.21.1 | Average Duration of VERVE Product Used per Use |
| Appendix | 16.2.6.21.2 | Total Duration of VERVE Product Used per Day |
| Appendix | 16.2.6.22 | Original and Factor Score to QSU-Brief Questionnaire |
| Appendix | 16.2.6.23.1 | Original Score to MCEQ Questionnaire |
| Appendix | 16.2.6.23.2 | Factor Score to MCEQ Questionnaire |
| Appendix | 16.2.6.24 | Use the Product Again Questionnaire |
| 16.2.7. | Individual | Adverse Event Listings |

| Appendix 16.2.7.1 | Adverse Events (I of II) |
|-------------------|---------------------------------------------|
| Appendix 16.2.7.2 | Adverse Events (II of II) |
| Appendix 16.2.7.3 | Adverse Event Preferred Term Classification |

# 16.2.8. Individual Laboratory Measurements and Other Safety Observations

| Appendix 16.2.8.1.1 | Clinical Laboratory Report - Serum Chemistry |
|----------------------|----------------------------------------------|
| Appendix 16.2.8.1.2 | Clinical Laboratory Report - Hematology |
| Appendix 16.2.8.1.3 | Clinical Laboratory Report - Urinalysis |
| Appendix 16.2.8.1.4 | Clinical Laboratory Report - Comments |
| Appendix 16.2.8.1.5 | Alcohol Breath Tests |
| Appendix 16.2.8.1.6 | Urine Drug Screens |
| Appendix 16.2.8.1.7 | Pregnancy Tests |
| Appendix 16.2.8.1.8 | FSH |
| Appendix 16.2.8.1.9 | Contraception |
| Appendix 16.2.8.1.10 | Urine Cotinine Screens |
| Appendix 16.2.8.1.11 | Serology Sample Collection |
| Appendix 16.2.8.2 | Vital Signs |
| Appendix 16.2.8.3 | 12-Lead Electrocardiogram |
| Appendix 16.2.8.4 | Smoking Cessation Information |

#### 12. TABLE SHELLS

The following table shells provide a framework for the display of data from this study. The shells may change due to unforeseen circumstances. These shells may not be reflective of every aspect of this study, but are intended to show the general layout of the tables that will be included in the final report.

Table 14.1.1.1 Summary of Disposition by Study Group and Overall

| | | Group | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Population | Category | Product -<br>Trial* | 1 | 2 | 3 | 4 | 5 | 6 | Overall# |
| Safety | Enrolled | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| - | Completed | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| | Discontinued Early | XX | XX | XX | XX | XX | XX | XX | XX |
| | <reason1></reason1> | XX | XX | XX | XX | XX | XX | XX | XX |
| | <reason2></reason2> | XX | XX | XX | XX | XX | XX | XX | XX |
| | <reason3></reason3> | XX | XX | XX | XX | XX | XX | XX | XX |
| mITT | Enrolled | | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| | Completed | | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| | Discontinued Early | | XX | XX | XX | XX | XX | XX | XX |
| | <reason1></reason1> | | XX | XX | XX | XX | XX | XX | XX |
| | <reason2></reason2> | | XX | XX | XX | XX | XX | XX | XX |
| | <reason3></reason3> | | XX | XX | XX | XX | XX | XX | XX |
| PP | Enrolled | | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| | Completed | | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| | Discontinued Early | | XX | XX | XX | XX | XX | XX | XX |
| | <reason1></reason1> | | XX | XX | XX | XX | XX | XX | XX |
| | <reason2></reason2> | | XX | XX | XX | XX | XX | XX | XX |
| | <reason3></reason3> | | XX | XX | XX | XX | XX | XX | XX |

Note: \* Only includes subjects that enrolled in the product trial period and dropped prior to randomization.
# Subjects who only participated in the product trial period are excluded from the Overall summary.

Group X = <description of groups>
mITT = Modified Intent-to-treat, PP = Per protocol

Program: /CAXXXXX/sas prg/stsas/PROGRAMNAME.SAS DDMMMYYYY HH:MM

Table 14.1.1.2 Summary of Disposition for Screen Failures

| Population | Category | |
|---|---|---|
| Screen Failuers | Screened Discontinued Early <reason1> <reason2> <reason3></reason3></reason2></reason1> | XXX<br>XX<br>XX<br>XX<br>XX |

Program: /CAXXXXX/sas\_prg/stsas/PROGRAMNAME.SAS DDMMMYYYY HH:MM

Table 14.1.2 Demographic Summary by Study Group and Overall

| | | | Product | | Group | | |
|---|---|---|---|---|---|---|---|
| Populati | on Trait | | Trial* | 1 | 2 | 6 | Overall# |
| Safety | Gender | Male<br>Female | X (XX.X%)<br>X (XX.X%) | X (XX.X%)<br>X (XX.X%) | X (XX.X%)<br>X (XX.X%) | X (XX.X%)<br>X (XX.X%) | X (XX.X%)<br>X (XX.X%) |
| | Race | XXXXXXXXX<br>XXXXX<br>XXXXX | X(XX.X%)<br>X(XX.X%)<br>X(XX.X%) | X(XX.X%)<br>X(XX.X%)<br>X(XX.X%) | X (XX.X%)<br>X (XX.X%)<br>X (XX.X%) | X (XX.X%)<br>X (XX.X%)<br>X (XX.X%) | X (XX.X%)<br>X (XX.X%)<br>X (XX.X%) |
| | Ethnicity | Hispanic or Latino<br>Not Hispanic or Latino | X (XX.X%)<br>X (XX.X%) | X (XX.X%)<br>X (XX.X%) | X (XX.X%)<br>X (XX.X%) | X (XX.X%)<br>X (XX.X%) | X (XX.X%)<br>X (XX.X%) |
| | Age (yrs) | n<br>Mean<br>SD<br>Minimum<br>Median<br>Maximum | X<br>X.X<br>X.XX<br>XX<br>XX | X<br>X.X<br>X.XX<br>XX<br>XX | X<br>X.X<br>X.XX<br>XX<br>XX<br>XX | X<br>X.X<br>X.XX<br>XX<br>X.X<br>XX | X<br>X.X<br>X.XX<br>XX<br>X.X<br>XX |

Note: \* Only includes subjects that enrolled in the product trial Period and dropped prior to randomization. # Subjects who only participated in the product trial period are excluded from the Overall summary.

Group X = <description of groups>

mITT = Modified Intent-to-treat, PP = Per protocol

Program: /CAXXXXX/sas prg/stsas/PROGRAMNAME.SAS DDMMMYYYY HH:MM

Programmer Note: Weight (kg), height (cm), BMI (kg/m^2), annual income and highest grade of school will also be included in the demographic summary table. mITT and PP population will also be presented.

Table 14.1.3 Smoking History by Study Group and Overall

| Population | Trait | | Product<br>Trial* | 1 | 2 | 6 | Overall# |
|---|---|---|---|---|---|---|---|
| Safety | CPD | n<br>Mean<br>SD<br>Minimum<br>Median<br>Maximum | X<br>X.X<br>X.XX<br>XX<br>X.X | X<br>X.X<br>X.XX<br>XX<br>XX<br>XX | X<br>X.X<br>X.XX<br>XX<br>XX<br>XX | X<br>X.X<br>X.XX<br>XX<br>XX<br>XX | X<br>X.X<br>X.XX<br>XX<br>XX<br>XX |
| | Years Smoked | n<br>Mean<br>SD<br>Minimum<br>Median<br>Maximum | X<br>X.X<br>X.XX<br>XX<br>X.X<br>XX | X<br>X.X<br>X.XX<br>XX<br>XX<br>XX | X<br>X.X<br>X.XX<br>XX<br>XX<br>XX | X<br>X.X<br>X.XX<br>XX<br>XX<br>X.X | X<br>X.X<br>X.XX<br>XX<br>XX<br>X.X |

Note: \* Only includes subjects that enrolled in the product trial Period and dropped prior to randomization.

# Subjects who only participated in the product trial period are excluded from the Overall summary.

CPD = Cigarettes per day

Group X = <description of groups>

mITT = Modified Intent-to-treat, PP = Per protocol

Program: /CAXXXXX/sas prg/stsas/PROGRAMNAME.SAS DDMMMYYYYY HH:MM

Programmer Note: Fagerstrom score will also be summarized in the table. mITT and PP population will also be presented.

Note: Summary Tables 14.2.1.1.1.1-2, 14.2.1.2.1.1-2, 14.2.1.3.1.1-2, 14.2.1.4.1.1-2, 14.2.1.5.1.1-2, 14.2.1.6.1.1-2, 14.2.1.7.1.1-2, 14.2.1.8.1.1-2, 14.2.1.9.1.1-2, 14.2.1.10.1.1-2, 14.2.1.11.1.1-2, 14.2.1.12.1.1-2, 14.2.1.13.1.1-2, 14.2.1.14.1.1-2, 14.2.1.15.1.1-2, 14.2.1.16.1.1-2, 14.2.1.17.1.1-2, 14.2.1.18.1.1-2, 14.2.1.19.1.1-2, and 14.2.1.20.1.1-2 will have the following format:

Page 1 of X Table 14.2.1.1.1.1 Summary of <Matrix> <Biomarker> (<units>) by Study Group and Study Day (<Population>)

| Studv Dav | Statistics | 1 | <br>2 | Group<br>3 | 4 | 5 | 6 |
|---|---|---|---|---|---|---|---|
| -1 | n | X | X | X | X | X | X |
| | n missing | X | X | X | X | X | X |
| | Mean | X.X | X.X | X.X | X.X | X <b>.</b> X | X.X |
| | SD | X.XX | X.XX | X.XX | X.XX | X.XX | X.XX |
| | CV (%) | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| | SEM | X.XX | X.XX | X.XX | X.XX | X.XX | X.XX |
| | Minimum | XX | XX | XX | XX | XX | XX |
| | Median | X.X | X.X | X.X | X.X | X.X | X.X |
| | Maximum | XX | XX | XX | XX | XX | XX |
| | 95% CI XX. | X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| 5 | n | X | X | X | X | X | X |
| | n missing | X | X | X | X | X | X |
| | Mean | X.X | X.X | X.X | X.X | X.X | X.X |
| | SD | X.XX | X.XX | X.XX | X.XX | X.XX | X.XX |
| | CV (%) | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| | SEM | X.XX | X.XX | X.XX | X.XX | X.XX | X.XX |
| | Minimum | XX | XX | XX | XX | XX | XX |
| | Median | X.X | X.X | X <b>.</b> X | X.X | X.X | X.X |
| | | XX | XX | XX | XX | XX | XX |
| | | | | | | XX.X, XX.X | |
| 7 | <same above<="" as="" td=""><td><b>&gt;</b></td><td></td><td></td><td></td><td></td><td></td></same> | <b>&gt;</b> | | | | | |

Group X = <description of groups>

Note: Summary tables 14.2.1.1.2.1-2, 14.2.1.2.2.1-2, 14.2.1.3.2.1-2, 14.2.1.4.2.1-2, 14.2.1.5.2.1-2, 14.2.1.6.2.1-2, 14.2.1.7.2.1-2, 14.2.1.8.2.1-2, 14.2.1.9.2.1-2, 14.2.1.10.2.1-2, 14.2.1.11.2.1-2, 14.2.1.12.2.1-2, 14.2.1.13.2.1-2, 14.2.1.14.2.1-2, 14.2.1.15.2.1-2, 14.2.1.16.2.1-2, 14.2.1.17.2.1-2, 14.2.1.18.2.1-2, 14.2.1.19.2.1-2, and 14.2.1.20.2.1-2 will have the following format:

| | Group Group | | | | | | |
|---|---|---|---|---|---|---|---|
| Study Day | Statistics | 1 | 2 | 3 | 4 | 5 | 6 |
| 5 | n | X | X | X | X | X | X |
| | n missing | X | X | X | X | X | X |
| | Mean | X.X | X.X | X.X | X.X | X.X | X.X |
| | SD | X.XX | X.XX | X.XX | X.XX | X.XX | X.XX |
| | CV (%) | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| | SEM | X.XX | X.XX | X.XX | X.XX | X.XX | X.XX |
| | Minimum | XX | XX | XX | XX | XX | XX |
| | Median | X.X | X.X | X.X | X.X | X.X | X.X |
| | Maximum | XX | XX | XX | XX | XX | XX |
| | 95% CI 2 | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| 7 | n | X | X | X | X | X | X |
| | n missing | X | X | X | X | X | X |
| | Mean | X.X | X.X | X.X | X.X | X.X | X.X |
| | SD | X.XX | X.XX | X.XX | X.XX | X.XX | X.XX |
| | CV (%) | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| | SEM | X.XX | X.XX | X.XX | X.XX | X.XX | X.XX |
| | Minimum | XX | XX | XX | XX | XX | XX |
| | Median | X.X | X.X | X.X | X.X | X.X | X.X |
| | Maximum | XX | XX | XX | XX | XX | XX |
| | 95% CI › | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |

\_\_\_\_\_

Baseline = Day -1

Group X = <description of groups>

Program: /CAXXXXX/sas prg/pksas/PROGRAMNAME.SAS DDMMMYYYY HH:MM

Table 14.2.1.1.3.1 Summary of <Matrix> <Biomarker> Percent Change from Baseline (%) by Study Group and Study Day (<Population>)

| | | | Group | | | | |
|---|---|---|---|---|---|---|---|
| Study Day | Statistics | 1 | 2 | 3 | 4 | 5 | 6 |
| 5 | n | X | X | X | X | X | X |
| | n missing | X | X | X | X | X | X |
| | Mean | X.X | X.X | X.X | X.X | X.X | X.X |
| | SD | X.XX | X.XX | X.XX | X.XX | X.XX | X.XX |
| | CV (%) | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| | SEM | X.XX | X.XX | X.XX | X.XX | X.XX | X.XX |
| | Minimum | XX | XX | XX | XX | XX | XX |
| | Median | X.X | X.X | X.X | X.X | X.X | X.X |
| | Maximum | XX | XX | XX | XX | XX | XX |
| | 95% CI X | XXX, XXX | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| 7 | n | X | X | X | Х | X | X |
| | n missing | X | X | X | X | X | X |
| | Mean | X.X | X.X | X.X | X.X | X.X | X.X |
| | SD | X.XX | X.XX | X.XX | X.XX | X.XX | X.XX |
| | CV (%) | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| | SEM | X.XX | X.XX | X.XX | X.XX | X.XX | X.XX |
| | Minimum | XX | XX | XX | XX | XX | XX |
| | Median | X.X | X.X | X.X | X.X | X.X | X.X |
| | Maximum | XX | XX | XX | XX | XX | XX |
| | | X.X, XX.X | XX.X, XX.X | | XX.X, XX.X | | XX.X, XX.X |

Baseline = Day -1

Group X = <description of groups>

Program: /CAXXXXX/sas\_prg/pksas/PROGRAMNAME.SAS DDMMMYYYY HH:MM

Note: Summary Tables 14.2.1.1.4.1-2, 14.2.1.2.4.1-2, 14.2.1.3.4.1-2, 14.2.1.4.4.1-2, 14.2.1.5.4.1-2, 14.2.1.6.4.1-2, 14.2.1.7.4.1-2, 14.2.1.8.4.1-2, 14.2.1.9.4.1-2, 14.2.1.10.4.1-2, 14.2.1.11.4.1-2, 14.2.1.12.4.1-2, 14.2.1.13.4.1-2, 14.2.1.14.4.1-2, 14.2.1.15.4.1-2, 14.2.1.16.4.1-2, 14.2.1.17.4.1-2, 14.2.1.18.4.1-2, and 14.2.1.19.4.1-2 will have the following format:

| Charles Dass | 04-44-44 | 1 | <br>2 | Group | 4 | <br>5 | · |
|---|---|---|---|---|---|---|---|
| Study Day<br> | Statistics | 1<br> | | 3 | 4<br> | ა<br> | b |
| -1 | n | X | X | X | X | X | X |
| | n missing | X | X | X | X | X | X |
| | Mean | X.X | X.X | X.X | X.X | X.X | X.X |
| | SD | X.XX | X.XX | X.XX | X.XX | X.XX | X.XX |
| | CV (%) | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| | SEM | X.XX | X.XX | X.XX | X.XX | X.XX | X.XX |
| | Minimum | XX | XX | XX | XX | XX | XX |
| | Median | X.X | X.X | X.X | X.X | X.X | X.X |
| | Maximum | XX | XX | XX | XX | XX | XX |
| | 95% CI XX. | X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| 5 | n | X | X | X | X | X | X |
| | n missing | X | X | X | X | X | X |
| | Mean | X.X | X.X | X.X | X.X | X.X | X.X |
| | SD | X.XX | X.XX | X.XX | X.XX | X.XX | X.XX |
| | CV (%) | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| | SEM | X.XX | X.XX | X.XX | X.XX | X.XX | X.XX |
| | Minimum | XX | XX | XX | XX | XX | XX |
| | Median | X.X | X.X | X.X | X.X | X.X | X.X |
| | Maximum | XX | XX | XX | XX | XX | XX |
| | 95% CI XX. | X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| 7 | <same above<="" as="" td=""><td><u>&gt;</u></td><td></td><td></td><td></td><td></td><td></td></same> | <u>&gt;</u> | | | | | |

Group X = <description of groups>

Program: /CAXXXXX/sas prg/pksas/PROGRAMNAME.SAS DDMMYYYYY HH:MM

Note: Statistical summary tables 14.2.1.1.5-6.1, 14.2.1.2.5-6.1, 14.2.1.3.5-6.1, 14.2.1.4.5-6.1, 14.2.1.5.5-6.1, 14.2.1.5.5-6.1, 14.2.1.1.5-6.1, 14.2.1.12.5-6.1, 14.2.1.13.5-6.1, 14.2.1.13.5-6.1, 14.2.1.13.5-6.1, 14.2.1.15.5-6.1, 14.2.1.16.5-6.1, 14.2.1.17.5-6.1, 14.2.1.18.5-6.1, 14.2.1.19.5-6.1, and 14.2.1.20.4-5.1 will have the following format:

Page 1 of X Table 14.2.1.1.5.1 Statistical Summary of <Matrix> <Biomarker>) (<Units>) by Study Group and Study Day (mITT Population)

| Group | Study Day | n | LS Mean | XX% Confidence Interval | p-value |
|-------|-----------|----|---------|-------------------------|---------|
| 1 | 5 | XX | X.XX | XX.XX - XXX.XX | X.XXXX |
| | 7 | XX | X.XX | XX.XX - XXX.XX | X.XXXX |
| 2 | 5 | XX | X.XX | XX.XX - XXX.XX | X.XXXX |
| | 7 | XX | X.XX | XX.XX - XXX.XX | X.XXXX |
| 3 | 5 | XX | X.XX | XX.XX - XXX.XX | X.XXXX |
| | 7 | XX | X.XX | XX.XX - XXX.XX | X.XXXX |
| 4 | 5 | XX | X.XX | XX.XX - XXX.XX | X.XXXX |
| | 7 | XX | X.XX | XX.XX - XXX.XX | X.XXXX |
| 5 | 5 | XX | X.XX | XX.XX - XXX.XX | X.XXXX |
| | 7 | XX | X.XX | XX.XX - XXX.XX | X.XXXX |
| 6 | 5 | XX | X.XX | XX.XX - XXX.XX | X.XXXX |
| | 7 | XX | X.XX | XX.XX - XXX.XX | X.XXXX |

Note: The mixed model for repeated measures includes study group, study day, study group by study visit interaction, and gender as fixed effects, baseline (Day -1)\_ value as the covariate with a variance-covariance matrix based on the AIC value. Final variance-covariance matrix is XXX.

n = Number of observation used in the analysis

Least-squares means (LS Means) are calculated from the MMRM.

Group  $X = \langle description \ of \ groups \rangle$ 

Program: /CAXXXXX/sas prg/pksas PROGRAMNAME.SAS DDMMMYYYY HH:MM

Note: Statistical Comparison tables 14.2.1.1.5-6.2, 14.2.1.2.5-6.2, 14.2.1.3.5-6.2, 14.2.1.4.5-6.2, 14.2.1.5.5-6.2, 14.2.1.5.5-6.2, 14.2.1.1.5-6.2, 14.2.1.12.5-6.2, 14.2.1.13.5-6.2, 14.2.1.13.5-6.2, 14.2.1.13.5-6.2, 14.2.1.13.5-6.2, 14.2.1.13.5-6.2, 14.2.1.15.5-6.2, 14.2.1.16.5-6.2, 14.2.1.17.5-6.2, 14.2.1.18.5-6.2, 14.2.1.19.5-6.2, and 14.2.1.20.4-5.2 will have the following format:

Page 1 of X Table 14.2.1.1.5.2 Statistical Comparisons of <Biomarker> (Units) Between Study Groups by Study Day (mITT Population)

| Comparison | Study Day | LS<br>Test (n) | S Means<br>Reference (n) | LS Mean Difference<br>(Test - Reference) | XX% Confidence Interval | p-value |
|---|---|---|---|---|---|---|
| Group 2 vs Group 1 | 5 | X.XX (X) | X.XX (X) | XXX.XX | xx.xx - xxx.xx | X.XXXX |
| | 7 | X.XX (X) | X.XX (X) | XXX.XX | XX.XX - XXX.XX | X.XXXX |
| Group 3 vs Group 1 | 5 | X.XX (X) | X.XX (X) | XXX.XX | XX.XX - XXX.XX | X.XXXX |
| | 7 | X.XX (X) | X.XX (X) | XXX.XX | XX.XX - XXX.XX | X.XXXX |
| Group 4 vs Group 1 | 5 | X.XX (X) | X.XX (X) | XXX.XX | XX.XX - XXX.XX | X.XXXX |
| | 7 | X.XX (X) | X.XX (X) | XXX.XX | XX.XX - XXX.XX | X.XXXX |
| Group 5 vs Group 1 | 5 | X.XX (X) | X.XX (X) | XXX.XX | XX.XX - XXX.XX | X.XXXX |
| | 7 | X.XX (X) | X.XX (X) | XXX.XX | XX.XX - XXX.XX | X.XXXX |
| Group 2 vs Group 6 | 5 | X.XX (X) | X.XX (X) | XXX.XX | xx.xx - xxx.xx | X.XXXX |
| | 7 | X.XX (X) | X.XX (X) | XXX.XX | XX.XX - XXX.XX | X.XXXX |
| Group 3 vs Group 6 | 5 | X.XX (X) | X.XX (X) | XXX.XX | XX.XX - XXX.XX | X.XXXX |
| | 7 | X.XX (X) | X.XX (X) | XXX.XX | XX.XX - XXX.XX | X.XXXX |
| Group 4 vs Group 6 | 5 | X.XX (X) | X.XX (X) | XXX.XX | XX.XX - XXX.XX | X.XXXX |
| | 7 | X.XX (X) | X.XX (X) | XXX.XX | XX.XX - XXX.XX | X.XXXX |
| Group 5 vs Group 6 | 5 | X.XX (X) | X.XX (X) | XXX.XX | XX.XX - XXX.XX | X.XXXX |
| | 7 | X.XX (X) | X.XX (X) | XXX.XX | XX.XX - XXX.XX | X.XXXX |

Note: The mixed model for repeated measures includes study group, study day, study group by study visit interaction, and gender as fixed effects, baseline (Day -1) value as the covariate with a variance-covariance matrix based on the AIC value.

Final variance-covariance matrix is XXX.

Test = The first group in the comparison

Reference = The second group in the comparison

n = Number of observation used in the analysis

Dunnett-Hsu adjusted confidence interval and p-value are reported.

Group  $X = \langle description \ of \ groups \rangle$ 

Program: /CAXXXXX/sas prg/pksas PROGRAMNAME.SAS DDMMMYYYY HH:MM

# Note: Statistical summary table 14.2.1.1.7.1 will have the following format:

Table 14.2.1.1.7.1 Statistical Summary of Total Urine NNAL 24-Hour Excreted (ng/24 hour) by Study Group (mITT Population with
Imputation of Missing Data Using Last Observation Carried Forward Method)

| Group | Study Day | n | LS Mean | XX% Confidence Interval | p-value |
|-------|-----------|----|---------|-------------------------|---------|
| 1 | 5 | XX | X.XX | XX.XX - XXX.XX | X.XXXX |
| | 7 | XX | X.XX | XX.XX - XXX.XX | X.XXXX |
| 2 | 5 | XX | X.XX | XX.XX - XXX.XX | X.XXXX |
| | 7 | XX | X.XX | XX.XX - XXX.XX | X.XXXX |
| 3 | 5 | XX | X.XX | XX.XX - XXX.XX | X.XXXX |
| | 7 | XX | X.XX | XX.XX - XXX.XX | X.XXXX |
| 4 | 5 | XX | X.XX | XX.XX - XXX.XX | X.XXXX |
| | 7 | XX | X.XX | XX.XX - XXX.XX | X.XXXX |
| 5 | 5 | XX | X.XX | XX.XX - XXX.XX | X.XXXX |
| | 7 | XX | X.XX | XX.XX - XXX.XX | X.XXXX |
| 6 | 5 | XX | X.XX | XX.XX - XXX.XX | X.XXXX |
| | 7 | XX | X.XX | XX.XX - XXX.XX | X.XXXX |

Note: The mixed model for repeated measures includes study group, study day, study group by study visit interaction, and gender as fixed effects, baseline (Day -1) value as the covariate with a variance-covariance matrix based on the AIC value. Final variance-covariance matrix is XXX.

n = Number of observation used in the analysis

Least-squares means (LS Means) are calculated from the MMRM.

Group  $X = \langle description \ of \ groups \rangle$ 

Program: /CAXXXXX/sas prg/pksas PROGRAMNAME.SAS DDMMYYYYY HH:MM

# Note: Statistical Comparison table 14.2.1.1.7.2 will have the following format:

Page 1 of X Table 14.2.1.1.7.2 Statistical Comparisons of Total Urine NNAL 24-Hour Excreted (ng/24 hour) Study Groups (mITT Population with Imputation of Missing Data Using Last Observation Carried Forward Method)

| Comparison | Study Day | LS<br>Test (n) | Means<br>Reference (n) | LS Mean Difference<br>(Test - Reference) | XX% Confidence Interval | p-value |
|---|---|---|---|---|---|---|
| Group 2 vs Group 1 | 5 | X.XX (X) | X.XX (X) | XXX.XX | xx.xx - xxx.xx | X.XXXX |
| | 7 | X.XX (X) | X.XX (X) | XXX.XX | XX.XX - XXX.XX | X.XXXX |
| Group 3 vs Group 1 | 5 | X.XX (X) | X.XX (X) | XXX.XX | XX.XX - XXX.XX | X.XXXX |
| | 7 | X.XX (X) | X.XX (X) | XXX.XX | XX.XX - XXX.XX | X.XXXX |
| Group 4 vs Group 1 | 5 | X.XX (X) | X.XX (X) | XXX.XX | XX.XX - XXX.XX | X.XXXX |
| | 7 | X.XX (X) | X.XX (X) | XXX.XX | XX.XX - XXX.XX | X.XXXX |
| Group 5 vs Group 1 | 5 | X.XX (X) | X.XX (X) | XXX.XX | XX.XX - XXX.XX | X.XXXX |
| | 7 | X.XX (X) | X.XX (X) | XXX.XX | XX.XX - XXX.XX | X.XXXX |
| Group 2 vs Group 6 | 5 | X.XX (X) | X.XX (X) | XXX.XX | xx.xx - xxx.xx | X.XXXX |
| | 7 | X.XX (X) | X.XX (X) | XXX.XX | XX.XX - XXX.XX | X.XXXX |
| Group 3 vs Group 6 | 5 | X.XX (X) | X.XX (X) | XXX.XX | XX.XX - XXX.XX | X.XXXX |
| | 7 | X.XX (X) | X.XX (X) | XXX.XX | XX.XX - XXX.XX | X.XXXX |
| Group 4 vs Group 6 | 5 | X.XX (X) | X.XX (X) | XXX.XX | XX.XX - XXX.XX | X.XXXX |
| | 7 | X.XX (X) | X.XX (X) | XXX.XX | XX.XX - XXX.XX | X.XXXX |
| Group 5 vs Group 6 | 5 | X.XX (X) | X.XX (X) | XXX.XX | XX.XX - XXX.XX | X.XXXX |
| | 7 | X.XX (X) | X.XX (X) | XXX.XX | xx.xx - xxx.xx | X.XXXX |

Note: The mixed model for repeated measures includes study group, study day, study group by study visit interaction, and gender as fixed effects, baseline (Day -1) value as the covariate with a variance-covariance matrix based on the AIC value.

Final variance-covariance matrix is XXX. Test = The first group in the comparison

Reference = The second group in the comparison

n = Number of observation used in the analysis

Dunnett-Hsu adjusted confidence interval and p-value are reported.

Group X = <description of groups>

Program: /CAXXXXX/sas prg/pksas PROGRAMNAME.SAS DDMMMYYYY HH:MM

# Note: Statistical summary table 14.2.1.1.8.1 will have the following format:

Page 1 of X Table 14.2.1.1.8.1 Statistical Summary of Total Urine NNAL 24-Hour Excreted (ng/24 hour) by Study Group (mITT Population with Imputation of Missing Data Using Multiple Imputation by SAS MI Procedure)

| Group | Study Day | n | LS Mean | - XX% Confidence Interval | p-value |
|-------|-----------|----|---------|---------------------------|---------|
| 1 | 7 | XX | X.XX | XX.XX - XXX.XX | X.XXXX |
| 2 | 7 | XX | X.XX | XX.XX - XXX.XX | X.XXXX |
| 3 | 7 | XX | X.XX | XX.XX - XXX.XX | X.XXXX |
| 4 | 7 | XX | X.XX | XX.XX - XXX.XX | X.XXXX |
| 5 | 7 | XX | X.XX | XX.XX - XXX.XX | X.XXXX |
| 6 | 7 | XX | X.XX | XX.XX - XXX.XX | X.XXXX |

Note: The mixed model includes study group and gender as fixed effects, and baseline (Day -1) value as the covariate. n = Number of observation used in the analysis Least-squares means (LS Means) are calculated from the ANCOVA.

Group X = <description of groups>

Program: /CAXXXX/sas prg/pksas PROGRAMNAME.SAS DDMMMYYYY HH:MM

# Note: Statistical Comparison table 14.2.1.1.8.2 will have the following format:

Table 14.2.1.1.8.2 Statistical Comparisons of Total Urine NNAL 24-Hour Excreted (ng/24 hour) Between Study Groups (mITT Population with Imputation of Missing Data Using Multiple Imputation by SAS MI Procedure)

| Comparison | Study Day | LS<br>Test (n) | Means Reference (n) | LS Mean Difference<br>(Test - Reference) | XX% Confidence Interval | p-value |
|---|---|---|---|---|---|---|
| Group 2 vs Group 1 | 7 | X.XX (X) | X.XX (X) | XXX.XX | XX.XX - XXX.XX | X.XXXX |
| Group 3 vs Group 1 | 7 | X.XX (X) | X.XX (X) | XXX.XX | XX.XX - XXX.XX | X.XXXX |
| Group 4 vs Group 1 | 7 | X.XX (X) | X.XX (X) | XXX.XX | XX.XX - XXX.XX | X.XXXX |
| Group 5 vs Group 1 | 7 | X.XX (X) | X.XX (X) | XXX.XX | XX.XX - XXX.XX | X.XXXX |
| Group 2 vs Group 6 | 7 | X.XX (X) | X.XX (X) | XXX.XX | XX.XX - XXX.XX | X.XXXX |
| Group 3 vs Group 6 | 7 | X.XX (X) | X.XX (X) | XXX.XX | XX.XX - XXX.XX | X.XXXX |
| Group 4 vs Group 6 | 7 | X.XX (X) | X.XX (X) | XXX.XX | XX.XX - XXX.XX | X.XXXX |
| Group 5 vs Group 6 | 7 | X.XX (X) | X.XX (X) | XXX.XX | XX.XX - XXX.XX | X.XXXX |

Note: The mixed model includes study group and gender as fixed effects, and baseline (Day -1) value as the covariate.

Least-squares means (LS Means) are calculated from the ANCOVA.

Test = The first group in the comparison

Reference = The second group in the comparison

n = Number of observation used in the analysis

Dunnett-Hsu adjusted confidence interval and p-value are reported.

Group X = <description of groups>

Program: /CAXXXXX/sas prg/pksas PROGRAMNAME.SAS DDMMMYYYY HH:MM

n = Number of observation used in the analysis

# Note: Summary Table 14.2.1.1.9.1 will have the following format:

| Study Day | Statistics | 1 | 2 | Group<br>3 | 4 | 5 | 6 |
|---|---|---|---|---|---|---|---|
| -1 | n | X | X | Х | X | X | X |
| | n missing | X | X | X | X | X | X |
| | Mean | X.X | X.X | X.X | X.X | X.X | X.X |
| | SD | X.XX | X.XX | X.XX | X.XX | X.XX | X.XX |
| | CV (%) | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| | SEM | X.XX | X.XX | X.XX | X.XX | X.XX | X.XX |
| | Minimum | XX | XX | XX | XX | XX | XX |
| | Median | X.X | X.X | X.X | X.X | X.X | X.X |
| | Maximum | XX | XX | XX | XX | XX | XX |
| | 95% CI XX | X.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| 5 | n | X | X | X | X | X | X |
| | n missing | X | X | X | X | X | X |
| | Mean | X.X | X.X | X.X | X.X | X.X | X.X |
| | SD | X.XX | X.XX | X.XX | X.XX | X.XX | X.XX |
| | CV (%) | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| | SEM | X.XX | X.XX | X.XX | X.XX | X.XX | X.XX |
| | Minimum | XX | XX | XX | XX | XX | XX |
| | Median | X.X | X.X | X.X | X.X | X.X | X.X |
| | Maximum | XX | XX | XX | XX | XX | XX |
| | 95% CI XX | X.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| 7 | <same abov<="" as="" td=""><td>7e&gt;</td><td></td><td></td><td></td><td></td><td></td></same> | 7e> | | | | | |

Group X = <description of groups>

Program: /CAXXXXX/sas\_prg/pksas/PROGRAMNAME.SAS DDMMMYYYY HH:MM

# Note: Statistical summary tables 14.2.1.1.9.2 and 14.2.1.1.10.1 will have the following format:

Page 1 of X Table 14.2.1.1.9.2 Statistical Summary of Total Urine NNAL 24-Hour Excreted (ng/24 hour) at Day 7 by Study Group (mITT Population with Outliers Excluded)

| Group | Study Day | n | LS Mean | XX% Confidence Interval | p-value |
|-------|-----------|----|---------|-------------------------|---------|
| 1 | 7 | XX | X.XX | XX.XX - XXX.XX | X.XXXX |
| 2 | 7 | XX | X.XX | XX.XX - XXX.XX | X.XXXX |
| 3 | 7 | XX | X.XX | XX.XX - XXX.XX | X.XXXX |
| 4 | 7 | XX | X.XX | XX.XX - XXX.XX | X.XXXX |
| 5 | 7 | XX | X.XX | XX.XX - XXX.XX | X.XXXX |
| 6 | 7 | XX | X.XX | XX.XX - XXX.XX | X.XXXX |

Note: The mixed model for repeated measures includes study group, study day, study group by study visit interaction, and gender as fixed effects, baseline (Day -1) value as the covariate with a variance-covariance matrix based on the AIC value. Final variance-covariance matrix is XXX.

n = Number of observation used in the analysis

Least-squares means (LS Means) are calculated from the MMRM.

Group X = <description of groups>

Program: /CAXXXXX/sas prg/pksas PROGRAMNAME.SAS DDMMMYYYY HH:MM

# Note: Statistical Comparison tables 14.2.1.1.9.3 and 14.2.1.1.10.2 will have the following format:

Table 14.2.1.1.9.3 Statistical Comparisons of Total Urine NNAL 24-Hour Excreted (ng/24 hour) at Day 7 Between Study Groups (mITT Population with Outliers Excluded)

| Comparison | Study Day | Test (n) | S Means<br>Reference (n) | LS Mean Difference<br>(Test - Reference) | XX% Confidence Interval | p-value |
|---|---|---|---|---|---|---|
| Group 2 vs Group 1 | 7 | X.XX (X) | X.XX (X) | XXX.XX | XX.XX - XXX.XX | X.XXXX |
| Group 3 vs Group 1 | 7 | X.XX (X) | X.XX (X) | XXX.XX | XX.XX - XXX.XX | X.XXXX |
| Group 4 vs Group 1 | 7 | X.XX (X) | X.XX (X) | XXX.XX | XX.XX - XXX.XX | X.XXXX |
| Group 5 vs Group 1 | 7 | X.XX (X) | X.XX (X) | XXX.XX | XX.XX - XXX.XX | X.XXXX |
| Group 2 vs Group 6 | 7 | X.XX (X) | X.XX (X) | XXX.XX | xx.xx - xxx.xx | X.XXXX |
| Group 3 vs Group 6 | 7 | X.XX (X) | X.XX (X) | XXX.XX | XX.XX - XXX.XX | X.XXXX |
| Group 4 vs Group 6 | 7 | X.XX (X) | X.XX (X) | XXX.XX | XX.XX - XXX.XX | X.XXXX |
| Group 5 vs Group 6 | 7 | X.XX (X) | X.XX (X) | XXX.XX | XX.XX - XXX.XX | X.XXXX |

Note: The mixed model for repeated measures includes study group, study day, study group by study visit interaction, and gender as fixed effects, baseline (Day -1) value as the covariate with a variance-covariance matrix based on the AIC value. Final variance-covariance matrix is XXX.

Least-squares means (LS Means) are calculated from the MMRM.

Test = The first group in the comparison

Reference = The second group in the comparison

n = Number of observation used in the analysis

Dunnett-Hsu adjusted confidence interval and p-value are reported.

Group X = <description of groups>

Program: /CAXXXXX/sas prg/pksas PROGRAMNAME.SAS DDMMMYYYY HH:MM

# Note: Summary table 14.2.2.1 will have the following format:

Table 14.2.2.1 Summary of Number of Cigarettes Smoked Per Day by Study Group and Study Day (mITT Population)

| | | | | | | Study I | Day | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Group | | -2 | -1 | Baseline | 1 | 2 | 3 | 4 | 5 | 6 | 7 |
| 1 | n | Х | Х | Х | X | Х | X | Х | Х | X | X |
| | n missing | X | X | X | X | X | X | X | X | X | X |
| | Mean | X.X | X.X | X.X | X.X | X.X | X.X | X.X | X.X | X.X | X.X |
| | SD | X.XX | X.XX | X.XX | X.XX | X.XX | X.XX | X.XX | X.XX | X.XX | X.XX |
| | CV (%) | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| | SEM | X.X | X.X | X.X | X.X | X.X | X.X | X.X | X.X | X.X | X.X |
| | Minimum | X | X | X | X | X | X | X | X | X | X |
| | Q1 | X.X | X.X | X.X | X.X | X.X | X.X | X.X | X.X | X.X | X.X |
| | Median | X | X | X | X | X | X | X | X | X | X |
| | Q3 | X.X | X.X | X.X | X.X | X.X | X.X | X.X | X.X | X.X | X.X |
| | Maximum | X.X | X.X | X.X | X.X | X.X | X.X | X.X | X.X | X.X | X.X |
| | 95% CI | X, X | X, $X$ | X, X | X, $X$ | X, $X$ | X, $X$ | X, $X$ | $X_{\prime}$ $X$ | X, $X$ | X, $X$ |

2 <same as above>

Note: Baseline = Average of Days -2 and -1.

Group X = <description of groups>

Program: /CAXXXXX/ECR/sas prg/pksas/PROGRAMNAME.sas DDMMYYYYY HH:MM

Programmer Note: Groups 2 through 6 will also be presented in the table. For groups 1, 2, and 3, there will be data for all study days (from Day -2 to Day 7). For Groups 4, 5, and 6, there will only have data for Days -2, -1, and baseline.

# Note: Summary tables 14.2.2.2, 14.2.2.3, and 14.2.2.4 will have the following format:

Page 1 of X Table 14.2.2.2 Summary of VERVE Product Used Per Day by Study Group and Study Day (mITT Population)

| | | | | Stu | idy Day - | | | |
|---|---|---|---|---|---|---|---|---|
| Group | | 1 | 2 | 3 | 4 | 5 | 6 | 7 |
| 2 | n | Х | X | X | X | X | X | X |
| | n missing | X | X | X | X | X | X | X |
| | Mean | X.X | X.X | X.X | X.X | X.X | X.X | X.X |
| | SD | X.XX | X.XX | X.XX | X.XX | X.XX | X.XX | X.XX |
| | CV (%) | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| | SEM | X.X | X.X | X.X | X.X | X.X | X.X | X.X |
| | Minimum | X | X | X | X | X | X | X |
| | Q1 | X.X | X.X | X.X | X.X | X.X | X.X | X.X |
| | Median | X | X | X | X | X | X | X |
| | Q3 | X.X | X.X | X.X | X.X | X.X | X.X | X.X |
| | Maximum | X.X | X.X | X.X | X.X | X.X | X.X | X.X |
| | 95% CI | X, X | X, X | X, X | X, X | X, X | X, X | X, X |
| 3 | <same above="" as=""></same> | | | | | | | |

Note: Group X = <description of groups>

Program: /CAXXXXX/ECR/sas prg/pksas/PROGRAMNAME.sas DDMMMYYYY HH:MM

Programmer Note: Groups 3, 4, and 5 will also be presented in the table.

# **QSU-Brief Questionnaire Summary Table 14.2.3.1.1 will have the following format:**

Table 14.2.3.1.1 Summary of QSU-Brief Factor Scores and Change from Pre Product Use by Study Group and Study Day (mITT Population)

| <question or<="" th=""><th></th><th></th><th></th><th></th><th></th><th> Gro</th><th>up</th><th></th><th></th></question> | | | | | | Gro | up | | |
|---|---|---|---|---|---|---|---|---|---|
| Subscale> | Study Day | Time Point | Statistics | 1 | 2 | 3 | 4 | 5 | 6 |
| XXXXX | -1 | Morning | n | X | X | Х | X | X | X |
| | | | n missing | X | X | X | X | X | X |
| | | | Mean | X.X | X.X | X.X | X.X | X.X | X.X |
| | | | SD | X.XX | X.XX | X.XX | X.XX | X.XX | X.XX |
| | | | CV (%) | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| | | | SEM | X.X | X.X | X.X | X.X | X.X | X.X |
| | | | Minimum | X | X | X | X | X | X |
| | | | Q1 | X.X | X.X | X.X | X.X | X.X | X.X |
| | | | Median | X.X | X.X | X.X | X.X | X.X | X.X |
| | | | Q3 | X.X | X.X | X.X | X.X | X.X | X.X |
| | | | Maximum | XX | XX | XX | XX | XX | XX |
| | | | 95% CI | X, $X$ | X, $X$ | X, $X$ | $X_{\prime}$ $X$ | $X_{\prime}$ $X$ | X, X |

Evening <Same as above>

Change <Same as above>

XXXXX <same for remaining questions or subscales>

\_\_\_\_\_\_

Note: Group X = <description of groups> Change = Evening score - Morning score

Program: /CAXXXXX/ECR/sas prg/pksas/PROGRAMNAME.sas DDMMYYYYY HH:MM

Programmer note: There are two factor score for QSU-Brief and the time points are Day -1 (morning and Evening), Day 1 (morning and Evening), Day 5 (morning and Evening), and Day 7 (morning and Evening).

# Note: Statistical summary table 14.2.3.1.2.1 will have the following format:

Table 14.2.3.1.2.1 Statistical Summary of QSU-Brief Factor Change from Pre Product Use Scores by Study Group and Study Day

(mITT Population)

| Factor | Group | Study Day | n | LS Mean | XX% Confidence Interval | p-value |
|---|---|---|---|---|---|---|
| 1 | 1 | 1<br>5<br>7 | XX<br>XX<br>XX | X.XX<br>X.XX<br>X.XX | XX.XX - XXX.XX<br>XX.XX - XXX.XX<br>XX.XX - XXX.XX | X.XXXX<br>X.XXXX<br>X.XXXX |
| | 2 | 1<br>5<br>7 | XX<br>XX<br>XX | X.XX<br>X.XX<br>X.XX | XX.XX - XXX.XX<br>XX.XX - XXX.XX<br>XX.XX - XXX.XX | X.XXXX<br>X.XXXX<br>X.XXXX |
| | 3 | 1<br>5<br>7 | XX<br>XX<br>XX | X.XX<br>X.XX<br>X.XX | XX.XX - XXX.XX<br>XX.XX - XXX.XX<br>XX.XX - XXX.XX | X.XXXX<br>X.XXXX<br>X.XXXX |

Note: The mixed model for repeated measures includes study group, study day, study group by study visit interaction, and gender as fixed effects, baseline (Day -1) value as the covariate with a variance-covariance matrix based on the AIC value. Final variance-covariance matrix is XXX.

n = Number of observation used in the analysis

Least-squares means (LS Means) are calculated from the MMRM.

Group X = <description of groups>

Program: /CAXXXX/sas prg/pksas PROGRAMNAME.SAS DDMMYYYY HH:MM

Programmer note: Groups 4-6 and Factor 2 will also be presented in the table.

# Note: Statistical Comparison table 14.2.3.1.2.2 will have the following format:

Table 14.2.3.1.2.2 Statistical Comparisons of QSU-Brief Factor Change from Pre Product Use Scores Between Study Groups by Study Day
(mITT Population)

| Factor | Comparison | Study Day | L:<br>Test (n) | S Means<br>Reference | | LS Mean Difference<br>(Test - Reference) | XX% Confidence Interval | p-value |
|---|---|---|---|---|---|---|---|---|
| 1 | Group 2 vs Group 1 | 1 | X.XX (X) | X.XX | (X) | XXX.XX | XX.XX - XXX.XX | X.XXXX |
| | | 5 | X.XX (X) | X.XX | (X) | XXX.XX | XX.XX - XXX.XX | X.XXXX |
| | | 7 | X.XX (X) | X.XX | (X) | XXX.XX | XX.XX - XXX.XX | X.XXXX |
| | Group 3 vs Group 1 | 1 | X.XX (X) | X.XX | (X) | XXX.XX | XX.XX - XXX.XX | X.XXXX |
| | | 5 | X.XX (X) | X.XX | (X) | XXX.XX | XX.XX - XXX.XX | X.XXXX |
| | | 7 | X.XX (X) | X.XX | (X) | XXX.XX | XX.XX - XXX.XX | X.XXXX |
| | Group 4 vs Group 1 | 1 | X.XX (X) | X.XX | (X) | XXX.XX | XX.XX - XXX.XX | X.XXXX |
| | - | 5 | X.XX (X) | X.XX | (X) | XXX.XX | XX.XX - XXX.XX | X.XXXX |
| | | 7 | X.XX (X) | X.XX | (X) | XXX.XX | XX.XX - XXX.XX | X.XXXX |
| | Group 5 vs Group 1 | 1 | X.XX (X) | X.XX | (X) | XXX.XX | XX.XX - XXX.XX | X.XXXX |
| | | 5 | X.XX (X) | X.XX | (X) | XXX.XX | XX.XX - XXX.XX | X.XXXX |
| | | 7 | X.XX (X) | X.XX | (X) | XXX.XX | XX.XX - XXX.XX | X.XXXX |

Note: The mixed model for repeated measures includes study group, study day, study group by study visit interaction, and gender as fixed effects, baseline (Day -1) value as the covariate with a variance-covariance matrix based on the AIC value.

Final variance-covariance matrix is XXX.

Test = The first group in the comparison

Reference = The second group in the comparison

n = Number of observation used in the analysis

Group  $X = \langle description \ of \ groups \rangle$ 

Program: /CAXXXXX/sas prg/pksas PROGRAMNAME.SAS DDMMMYYYY HH:MM

Programmer note: Comparisons for Groups 2-5 versus Group 6 and Factor 2 will also be presented in the table.

# mCEQ Questionnaire Summary Table 14.2.3.1.1 will have the following format:

Table 14.2.3.2.1 Summary of mCEQ Factor Scores by Study Group and Study Day (mITT Population)

| Question or | | | | | | Gro | up | | |
|---|---|---|---|---|---|---|---|---|---|
| Subscale> | Study Day | Questionnaire | Statistics | 1 | 2 | 3 | 4 | 5 | 6 |
| XXXXX | -1 | mCEQ-C | n | X | Х | Х | Х | Х | X |
| | | | n missing | X | X | X | X | X | X |
| | | | Mean | X.X | X.X | X.X | X.X | X.X | X.X |
| | | | SD | X.XX | X.XX | X.XX | X.XX | X.XX | X.XX |
| | | | CV (%) | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| | | | SEM | X.X | X.X | X.X | X.X | X.X | X.X |
| | | | Minimum | X | X | X | X | X | X |
| | | | Q1 | X.X | X.X | X.X | X.X | X.X | X.X |
| | | | Median | X.X | X.X | X.X | X.X | X.X | X.X |
| | | | Q3 | X.X | X.X | X.X | X.X | X.X | X.X |
| | | | Maximum | XX | XX | XX | XX | XX | XX |
| | | | 95% CI | X, X | X, X | X, X | X, X | X, X | X, X |
| | 1 | mCEQ-C < | :Same as above> | | | | | | |

Note: Group X = <description of groups>

Program: /CAXXXX/ECR/sas prg/pksas/PROGRAMNAME.sas DDMMYYYYY HH:MM

Programmer note: There are five factor scores for mCEQ and the time points are Day -1, Day 1, Day 5, and Day 7. On Day -1, all groups have the values for mCEQ-C. For Group 1, mCEQ-C will be used for Days 1, 5, and 7. For Groups 2 and 3, both mCEQ-C and mCEQ-V will be used for Days 1, 5, and 7. For Groups 4 and 5, mCEQ-V will be used for Days 1, 5, and 7. No mCEQ for Group 6 after Day 1.

# Note: Statistical summary table 14.2.3.2.2.1 will have the following format:

Table 14.2.3.2.2.1 Statistical Summary of MCEQ-C Factor Scores by Study Group and Study Day

(mITT Population)

| Factor | Group | Study Day | n | LS Mean | XX% Confidence Interval | p-value |
|---|---|---|---|---|---|---|
| XXX | 1 | 1<br>5<br>7 | XX<br>XX<br>XX | X.XX<br>X.XX<br>X.XX | XX.XX - XXX.XX<br>XX.XX - XXX.XX<br>XX.XX - XXX.XX | X.XXXX<br>X.XXXX<br>X.XXXX |
| | 2 | 1<br>5<br>7 | XX<br>XX<br>XX | X.XX<br>X.XX<br>X.XX | XX.XX - XXX.XX<br>XX.XX - XXX.XX<br>XX.XX - XXX.XX | X.XXXX<br>X.XXXX<br>X.XXXX |
| | 3 | 1<br>5<br>7 | XX<br>XX<br>XX | X.XX<br>X.XX<br>X.XX | XX.XX - XXX.XX<br>XX.XX - XXX.XX<br>XX.XX - XXX.XX | X.XXXX<br>X.XXXX<br>X.XXXX |

Note: The mixed model for repeated measures includes study group, study day, study group by study visit interaction, and gender as fixed effects, baseline (Day -1) value as the covariate with a variance-covariance matrix based on the AIC value. Final variance-covariance matrix is XXX.

n = Number of observation used in the analysis

Least-squares means (LS Means) are calculated from the MMRM.

Group X = <description of groups>

Program: /CAXXXX/sas prg/pksas PROGRAMNAME.SAS DDMMMYYYY HH:MM

Programmer note: All factor scores will be presented in the table. This analysis only contains data from Groups 1-3.

# Note: Statistical Comparison table 14.2.3.2.2.2 will have the following format:

Table 14.2.3.2.2.2 Statistical Comparisons of mCEQ-C Factor Scores Between Study Groups by Study Day (mITT Population)

| | | | L | S Means | | LS Mean Difference | | |
|---|---|---|---|---|---|---|---|---|
| Factor | Comparison | Study Day | Test (n) | Reference ( | (n) | (Test - Reference) | XX% Confidence Interval | p-value |
| XXX | Group 2 vs Group 1 | 1 | X.XX (X) | X.XX ( | (X) | XXX.XX | XX.XX - XXX.XX | X.XXXX |
| | | 5 | X.XX (X) | X.XX ( | (X) | XXX.XX | XX.XX - XXX.XX | X.XXXX |
| | | 7 | X.XX (X) | X.XX ( | (X) | XXX.XX | XX.XX - XXX.XX | X.XXXX |
| | Group 3 vs Group 1 | 1 | X.XX (X) | X.XX ( | (X) | XXX.XX | XX.XX - XXX.XX | X.XXXX |
| | - | 5 | X.XX (X) | X.XX ( | (X) | XXX.XX | XX.XX - XXX.XX | X.XXXX |
| | | 7 | X.XX (X) | X.XX ( | (X) | XXX.XXX | XX.XX - XXX.XX | X.XXXX |

Note: The mixed model for repeated measures includes study group, study day, study group by study visit interaction, and gender as fixed effects, baseline (Day -1) value as the covariate with a variance-covariance matrix based on the AIC value.

Final variance-covariance matrix is XXX. Test = The first group in the comparison

Reference = The second group in the comparison

n = Number of observation used in the analysis

Group X = <description of groups>

Program: /CAXXXXX/sas prg/pksas PROGRAMNAME.SAS DDMMMYYYY HH:MM

Programmer note: Comparisons for all factor scores will also be presented in the table. This analysis only contains data from Groups 1-3.

# Note: Statistical summary table 14.2.3.2.3.1 will have the following format:

Table 14.2.3.2.3.1 Statistical Summary of MCEQ-V Factor Scores by Study Group and Study Day

(mITT Population)

| Factor | Group | Study Day | n | LS Mean | XX% Confidence Interval | p-value |
|---|---|---|---|---|---|---|
| XXX | 2 | 1<br>5<br>7 | XX<br>XX<br>XX | X.XX<br>X.XX<br>X.XX | XX.XX - XXX.XX<br>XX.XX - XXX.XX<br>XX.XX - XXX.XX | X.XXXX<br>X.XXXX<br>X.XXXX |
| | 3 | 1<br>5<br>7 | XX<br>XX<br>XX | X.XX<br>X.XX<br>X.XX | XX.XX - XXX.XX<br>XX.XX - XXX.XX<br>XX.XX - XXX.XX | X.XXXX<br>X.XXXX<br>X.XXXX |
| | 4 | 1<br>5<br>7 | XX<br>XX<br>XX | X.XX<br>X.XX<br>X.XX | XX.XX - XXX.XX<br>XX.XX - XXX.XX<br>XX.XX - XXX.XX | X.XXXX<br>X.XXXX<br>X.XXXX |
| | 5 | 1<br>5<br>7 | XX<br>XX<br>XX | X.XX<br>X.XX<br>X.XX | XX.XX - XXX.XX<br>XX.XX - XXX.XX<br>XX.XX - XXX.XX | X.XXXX<br>X.XXXX<br>X.XXXX |

Note: The mixed model for repeated measures includes study group, study day, study group by study visit interaction, and gender as fixed effects, baseline (Day -1) value as the covariate with a variance-covariance matrix based on the AIC value. Final variance-covariance matrix is XXX.

n = Number of observation used in the analysis

Least-squares means (LS Means) are calculated from the MMRM.

Group X = <description of groups>

Program: /CAXXXXX/sas prg/pksas PROGRAMNAME.SAS DDMMMYYYY HH:MM

Programmer note: All factor scores will be presented in the table. This analysis only contains data from Groups 2-5.

# Note: Statistical Comparison table 14.2.3.2.2.2 will have the following format:

Table 14.2.3.2.2.2 Statistical Comparisons of mCEQ-C Factor Scores Between Study Groups by Study Day (mITT Population)

| | | | L: | S Means | | LS Mean Difference | | |
|---|---|---|---|---|---|---|---|---|
| Factor | Comparison | Study Day | Test (n) | Reference ( | n) | (Test - Reference) | XX% Confidence Interval | p-value |
| XXX | Group 2 vs Group 4 | 1 | X.XX (X) | X.XX ( | X) | XXX.XX | xx.xx - xxx.xx | X.XXXX |
| | | 5 | X.XX (X) | X.XX ( | X) | XXX.XX | XX.XX - XXX.XX | X.XXXX |
| | | 7 | X.XX (X) | X.XX ( | X) | XXX.XX | XX.XX - XXX.XX | X.XXXX |
| | Group 3 vs Group 5 | 1 | X.XX (X) | X.XX ( | X) | XXX.XX | XX.XX - XXX.XX | X.XXXX |
| | - | 5 | X.XX (X) | X.XX ( | X) | XXX.XX | XX.XX - XXX.XX | X.XXXX |
| | | 7 | X.XX (X) | X.XX ( | X) | XXX.XX | XX.XX - XXX.XX | X.XXXX |

Note: The mixed model for repeated measures includes study group, study day, study group by study visit interaction, and gender as fixed effects, baseline (Day -1) value as the covariate with a variance-covariance matrix based on the AIC value.

Final variance-covariance matrix is XXX. Test = The first group in the comparison

Reference = The second group in the comparison

n = Number of observation used in the analysis

Group X = <description of groups>

Program: /CAXXXXX/sas prg/pksas PROGRAMNAME.SAS DDMMMYYYY HH:MM

Programmer note: Comparisons for all factor scores will also be presented in the table. This analysis only contains data from Groups 2-5.

# **Use Product Again Questionnaire Frequency Count Table 14.2.3.3.1 will have the following format:**

Table 14.2.3.3.1 Frequency of Response to Use the Product Again VAS Scores by Study Group and Study Product
(mITT Population)

| Question | Group | Statistics | -50 to <0 | 0 | >0 to 50 |
|---|---|---|---|---|---|
| Use Cigarette Again | 1 | n (%)<br>n (%) | XX (XX%)<br>XX (XX%) | XX (XX%)<br>XX (XX%) | XX (XX%)<br>XX (XX%) |
| | 2 | n (%)<br>n (%) | XX (XX%)<br>XX (XX%) | XX (XX%)<br>XX (XX%) | XX (XX%)<br>XX (XX%) |
| | 3 | n (%)<br>n (%) | XX (XX%)<br>XX (XX%) | XX (XX%)<br>XX (XX%) | XX (XX%)<br>XX (XX%) |
| Use VERVE Again | 2 | n (%)<br>n (%) | XX (XX%)<br>XX (XX%) | XX (XX%)<br>XX (XX%) | XX (XX%)<br>XX (XX%) |
| | 3 | n (%)<br>n (%) | XX (XX%)<br>XX (XX%) | XX (XX%)<br>XX (XX%) | XX (XX%)<br>XX (XX%) |
| | 4 | n (%)<br>n (%) | XX (XX%)<br>XX (XX%) | XX (XX%)<br>XX (XX%) | XX (XX%)<br>XX (XX%) |
| | 5 | n (응)<br>n (응) | XX (XX%)<br>XX (XX%) | XX (XX%)<br>XX (XX%) | XX (XX%)<br>XX (XX%) |

Note: Group X = <description of groups>

Program: /CAXXXXX/sas prg/pksas/PROGRAMNAME.SAS DDMMYYYYY HH:MM

Programmer note: Use product again for cigarettes will be presented for Groups 1 – 3. Use product again for VERVE will be presented for Groups 2, 3, 4 and 5. The questionnaire will not be conducted for Group 6.

# Use Product Again Questionnaire Summary Table 14.2.3.3.2 will have the following format:

Summary of Use Product Again Scores by Study Group and Study Product (mITT Population) Table 14.2.3.3.2

| | | | | Grou | 0 | |
|---|---|---|---|---|---|---|
| Product | Statistics | 1 | 2 | 3 | 4 | 5 |
| <br>Cigarette | n | Х | X | Х | | |
| | n missing | X | X | X | | |
| | Mean | X.X | X.X | X.X | | |
| | SD | X.XX | X.XX | X.XX | | |
| | CV (%) | XX.X | XX.X | XX.X | | |
| | SEM | X.X | X.X | X.X | | |
| | Minimum | X | X | X | | |
| | Q1 | X.X | X.X | X.X | | |
| | Median | X.X | X.X | X.X | | |
| | Q3 | X.X | X.X | X.X | | |
| | Maximum | XX | XX | XX | | |
| | 95% CI | X, X | X, X | X, X | | |
| VERVE | <same abov<="" as="" td=""><td>7e&gt;</td><td></td><td></td><td></td><td></td></same> | 7e> | | | | |

Note: Group X = <description of groups>

Program: /CAXXXXX/ECR/sas prg/pksas/PROGRAMNAME.sas DDMMMYYYY HH:MM

Programmer note: Use product again for cigarettes will be presented for Groups 1 – 3. Use product again for VERVE will be presented for Groups 2, 3, 4 and 5. The questionnaire will not be conducted for Group 6.

# Use Product Again Questionnaire Summary Table 14.2.3.3.3 will have the following format:

Table 14.2.3.3.3 Summary of Response to Use the Product Again Bipolar Scores by Category, Study Group and Study Product (mITT Population)

| Product Cigarette | Statistics<br><br>n | 1 | | 2 | | 3 | | 4 | į |
|---|---|---|---|---|---|---|---|---|---|
| | | -50 to < | <0 >0 to 50 | -50 to < | 0 >0 to 50 | -50 to < | ) >0 to 50 | | |
| | | Х | Х | Х | X | Х | X | | |
| | Mean | X.X | X.X | X.X | X.X | X.X | X.X | | |
| | SD | X.XX | X.XX | X.XX | X.XX | X.XX | X.XX | | |
| | CV(%) | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | | |
| | SEM | X.X | X.X | X.X | X.X | X.X | X.X | | |
| | Minimum | X | X | X | X | X | X | | |
| | Q1 | X.X | X.X | X.X | X.X | X.X | X.X | | |
| | Median | X.X | X.X | X.X | X.X | X.X | X.X | | |
| | Q3 | X.X | X.X | X.X | X.X | X.X | X.X | | |
| | Maximum | XX | XX | XX | XX | XX | XX | | |
| | 95% CI | X, X | X, X | X, X | X, X | X, X | X, X | | |

\_\_\_\_\_\_

Note: Group X = <description of groups>

Program: /CAXXXXX/ECR/sas prg/pksas/PROGRAMNAME.sas DDMMMYYYY HH:MM

Programmer note: Use product again for cigarettes will be presented for Groups 1 – 3. Use product again for VERVE will be presented for Groups 2, 3, 4 and 5. The questionnaire will not be conducted for Group 6.

Table 14.3.1.1 Adverse Event Frequency by Study Group - Number of Subjects Reporting the Event (% of Subjects Who Received Study Product Or in a Study group)

| | December 1 | | | | |
|---|---|---|---|---|---|
| Adverse Event* | Product<br>Trial\$ | 1 | 2 | . 6 | Overall# |
| Number of Subjects Who Received Study Product Or in a Study Group | XX (100%) | XX (100%) | XX (100%) | XX (100%) | XX (100%) |
| Number of Subjects With Adverse Events | X( X%) | X( X%) | X( XX%) | X( X%) | X( X%) |
| Number of Subjects Without Adverse Events | XX(XXX%) | XX(XX%) | XX(XX%) | XX(XX%) | XX (XXX%) |
| Eye disorders | X( X%) | X( X%) | X( X%) | X ( X%) | X( X%) |
| Vision blurred | X( X%) | X(X%) | X( X%) | X( X%) | X(X%) |
| Gastrointestinal disorders | X( X%) | X(X%) | X(X%) | X(X%) | X(X%) |
| Dyspepsia | X( X%) | X(X%) | X(X%) | X(X%) | X(X%) |
| Nausea | X( X%) | X(X%) | X(X%) | X(X%) | X(X%) |
| Musculoskeletal and connective tissue | X( X%) | X( X%) | X(X%) | X(X%) | X(X%) |
| disorders | | | | | |
| Back pain | X(X%) | X( X%) | X(X%) | X(X%) | X(X%) |
| Muscle cramps | X(X%) | X( X%) | X(X%) | X(X%) | X(X%) |
| Musculoskeletal pain | X( X%) | X(X%) | X( X%) | X( X%) | X( X%) |
| Nervous system disorders | X( X%) | X(X%) | X( X%) | X( X%) | X( X%) |
| Headache NOS | X( X%) | X(X%) | X( X%) | X( X%) | X( X%) |
| Reproductive system and breast disorders | X( X%) | X(X%) | X( X%) | X( X%) | X( X%) |
| Vaginal discharge | X( X%) | X(X%) | X(X%) | X(X%) | X(X%) |
| Respiratory, thoracic and mediastinal | X( X%) | X(X%) | X(X%) | X(X%) | X(X%) |
| disorders | | | | | |
| Epistaxis | X( X%) | X( X%) | X( X%) | X( X%) | X( X%) |

Note:  $\star$  Adverse events are classified according to MedDRA Version 20.0.

Group  $X = \langle description \ of \ groups \rangle$ 

Program: /CAXXXXX/sas prg/stsas/tab cdash tblae1a auto.sas DDMMMYYYYY HH:MM

<sup>\$</sup> Only includes adverse events that occurred during the product trial period.

<sup>#</sup> Adverse events that occurred during the product trial period are excluded from the Overall summary.
Table 14.3.1.2 Adverse Event Frequency by Study Group Number of Adverse Events (% of Total Adverse Events)

C----

| | Donalous | | | | |
|---|---|---|---|---|---|
| Adverse Event* | Product<br>Trial\$ | 1 | 2 | 6 | Overall# |
| Number of Adverse Events | XX (100%) | XX (100%) | XX(100%) | XX(100%) | XX (100%) |
| Eye disorders Vision blurred Gastrointestinal disorders Dyspepsia Nausea Musculoskeletal and connective tissue disorders Back pain Muscle cramps Musculoskeletal pain Nervous system disorders Headache NOS Reproductive system and breast disorders Vaginal discharge | X( X%) | X( X%) | X( X%) | X( X%) | X( X%) |
| Respiratory, thoracic and mediastinal disorders Epistaxis | X ( X%)<br>X ( X%) | X ( X%) | X ( X%)<br>X ( X%)<br>X ( X%) | X ( X%)<br>X ( X%) | X ( X%)<br>X ( X%)<br>X ( X%) |

Note: \* Adverse events are classified according to MedDRA Version 20.0.

Group X = <description of groups>

Program: /CAXXXXX/sas prg/stsas/tab cdash tblaela auto.sas DDMMMYYYY HH:MM

<sup>\$</sup> Only includes adverse events that occurred during the product trial period.

<sup>#</sup> Adverse events that occurred during the product trial period are excluded from the Overall summary.


| Table 14.3.1.3 | Adverse Event Frequency by | Study Product, Severity, | and Relationship to Study Group |
|---|---|---|---|
| | - Number of | Subjects Reporting Event | S |

| | | Number of<br>Subjects with | | Sever | ity | Relat | ionship to | Study Pro | duct | |
|---|---|---|---|---|---|---|---|---|---|---|
| Adverse Event* | Group | Adverse Events | Mild | Moderate | Severe | Not Related | Unlikely | Possibly | Likely | Definitely |
| Abdominal pain<br>Constipation<br>Dry throat<br>Headache | X<br>X<br>Product Tria<br>X | X<br>X<br>X<br>X | X<br>X<br>X<br>X | X<br>X<br>X<br>X | X<br>X<br>X | X<br>X<br>X<br>X | X<br>X<br>X<br>X | X<br>X<br>X<br>X | X<br>X<br>X<br>X | X<br>X<br>X<br>X |
| Product trial\$ Group 1 Group 2 Group 3 Group 4 Group 5 Group 6 Overall# | | X<br>X<br>X<br>X<br>X<br>X<br>X | X<br>X<br>X<br>X<br>X<br>X<br>X | X<br>X<br>X<br>X<br>X<br>X<br>X | X<br>X<br>X<br>X<br>X<br>X<br>X | X<br>X<br>X<br>X<br>X<br>X<br>X | X<br>X<br>X<br>X<br>X<br>X<br>X | X<br>X<br>X<br>X<br>X<br>X<br>X | X<br>X<br>X<br>X<br>X<br>X<br>X | X<br>X<br>X<br>X<br>X<br>X<br>X |

Note: \* Adverse events are classified according to MedDRA Version 20.0.

When a subject experienced the same AE at more than one level of severity during a product use period, only the most severe occurrence was counted.

When a subject experienced the same AE at more than one level of product relationship during a product use period, only the occurrence most closely related to study product was counted.

Group X = <description of groups>

Program: /CAXXXXX/sas prg/stsas/tab cdash tblae3a auto.sas DDMMMYYYY HH:MM

<sup>\$</sup> Only includes adverse events that occurred during the product trial period.

<sup>#</sup> Adverse events that occurred during the product trial period are excluded from the Overall summary.

Table 14.3.1.4 Adverse Event Frequency by Study Product, Severity, and Relationship to Study Group - Number of Adverse Events

| | | Novele and a G | Severity | | | Relationship to Study Product | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Adverse Event* | Group | Number of<br>Adverse Events | Mild | Moderate | Severe | Not Related | Unlikely | Possibly | Likely | Definitely |
| Abdominal pain | X | X | Х | X | Х | X | Х | Х | Х | X |
| Constipation | X | X | X | X | X | X | X | X | X | X |
| Dry throat | Product trial | X | X | X | X | X | X | X | X | X |
| Headache | X | X | X | X | X | X | X | X | X | X |
| Product trial\$ | | X | Х | X | Х | X | Х | X | Х | X |
| Group 1 | | X | X | X | X | X | X | X | X | X |
| Group 2 | | X | X | X | X | X | X | X | X | X |
| Group 3 | | X | X | X | X | X | X | X | X | X |
| Group 4 | | X | X | X | X | X | X | X | X | X |
| Group 5 | | X | X | X | X | X | X | X | X | X |
| Group 6 | | X | X | X | X | X | X | X | X | X |
| Overall# | | X | X | X | X | X | X | X | X | X |

Note: \* Adverse events are classified according to MedDRA Version 20.0.

Group  $X = \langle description \ of \ groups \rangle$ 

Program: /CAXXXXX/sas prg/stsas/tab cdash tblae4a auto.sas DDMMMYYYY HH:MM

<sup>\$</sup> Only includes adverse events that occurred during the product trial period.
# Adverse events that occurred during the product trial period are excluded from the Overall summary.


Table 14.3.2.1 Serious Adverse Events

\_\_\_\_\_

There were no serious adverse events recorded during the study

Program: /CAXXXXX/sas\_prg/stsas/tab cdash\_tblae\_ser.sas DDMMMYYYY HH:MM


Table 14.3.4.1 Out-of-Range Values and Recheck Results - Serum Chemistry

| Subject | Age/ | Study Visit | | | Parameter1 | Parameter2 | Parameter3 | Parameter4 | Parameter5 |
|---|---|---|---|---|---|---|---|---|---|
| Site Number | Gender | Name | Date | Group | | | | | |
| XXX XXXXXX | XX/X | Screenin | ng DDMMYYYY<br>DDMMYYYYY | × | XX HN<br>XX HN | XX LN<br>XX LN | XX<br>XX | XX<br>XX | XX HN<br>XX HN |

Note: Refer to Appendix 16.1.10.1 for the reference ranges of clinical laboratory tests.

 ${\tt H} = {\tt Above}$  Reference Range, L = Below Reference Range PI Interpretation: N = Not Clinically Significant

Group X = <description of groups>

Program: /CAXXXXX/sas prg/stsas/lis PROGRAMNAME.sas DDMMMYYYY HH:MM

Programmer Note: In the shell above, replace Parameter1, 2 etc. with actual lab tests in the study. Table 14.3.4.2 (hematology) and Table 14.3.4.3 (Urinalysis) will resemble Table 14.3.4.1.

Table 14.3.5.1 Clinical Laboratory Summary - Serum Chemistry

| | | | | | | Group | | |
|---|---|---|---|---|---|---|---|---|
| Laboratory Test (units) | Normal<br>Range | Time Point | Statistic | Product<br>Trial\$ | 1 | 2 | <b>.</b> 6 | Overall* |
| Testname (unit) | < - > | Screening | n | X | X | X | X | X |
| | | - | Mean | X.X | X.X | X.X | X.X | X.X |
| | | | SD | X.XX | X.XX | X.XX | X.XX | X.XX |
| | | | Minimum | XX | XX | XX | XX | XX |
| | | | Median | X.X | X.X | X.X | X.X | X.X |
| | | | Maximum | XX | XX | XX | XX | XX |
| | | End-of-Study | n | X | X | X | X | X |
| | | - | Mean | X.X | X.X | X.X | X.X | X.X |
| | | | SD | X.XX | X.XX | X.XX | X.XX | X.XX |
| | | | Minimum | XX | XX | XX | XX | XX |
| | | | Median | X.X | X.X | X . X | X.X | X.X |
| | | | Maximum | XX | XX | XX | XX | XX |

Note: # = Lowest of the lower ranges and highest of the higher ranges are used. Refer to Appendix 16.1.10.1 for the breakdown.

Group  $X = \langle description \ of \ groups \rangle$ 

Program: /CAXXXXX/sas\_prg/stsas/tab cdash\_labsummary.sas DDMMMYYYY HH:MM

Programmer Note: Tables 14.3.5.2 (hematology summary), 14.3.5.3 (urinalysis summary) will resemble 14.3.5.1.

<sup>\$</sup> Includes subjects only attended the product trial period.

<sup>\*</sup> Subjects only attended the product trial period are excluded from overall summarization.

Table 14.3.5.4 Vital Sign Summary

| | | | Droduct | | | | |
|---|---|---|---|---|---|---|---|
| Vital Sign (units) | Time Point | Statistic | Product<br>Trial\$ | 1 | 2 | 6 | Overall* |
| Testname (unit) | Screening | n | X | Х | X | X | Х |
| | | Mean | X.X | X.X | X.X | X.X | X.X |
| | | SD | X.XX | X.XX | X.XX | X.XX | X.XX |
| | | Minimum | XX | XX | XX | XX | XX |
| | | Median | X.X | X.X | X.X | X.X | X.X |
| | | Maximum | XX | XX | XX | XX | XX |
| | XXXXX | n | X | X | X | X | X |
| | | Mean | X.X | X.X | X.X | X.X | X.X |
| | | SD | X.XX | X.XX | X.XX | X.XX | X.XX |
| | | Minimum | XX | XX | XX | XX | XX |
| | | Median | X.X | X.X | X.X | X.X | X.X |
| | | Maximum | XX | XX | XX | XX | XX |
| | XXXXXX | n | | X | X | X | X |
| | | Mean | | X.X | X.X | X.X | X.X |
| | | SD | | X.XX | X.XX | X.XX | X.XX |
| | | Minimum | | XX | XX | XX | XX |
| | | Median | | X.X | X.X | X.X | X.X |
| | | Maximum | | XX | XX | XX | XX |

Group X = <description of groups>

Program: /CAXXXXX/sas prg/stsas/tab cdash vitsummary.sas DDMMMYYYY HH:MM

Programmer Note: In the shell above, replace Testname with actual variables in the study. Data will also be reported for Screening, Check-in, and End-of-Study.

Note: \$ Includes subjects only attended the product trial period.

\* Subjects only attended the product trial period are excluded from overall summarization.

### 13. LISTING SHELLS

The following listing shells provide a framework for the display of data from this study. The shells may change due to unforeseen circumstances. These shells may not be reflective of every aspect of this study, but are intended to show the general layout of the listings that will be included in the final report.

Note: Subjects only enrolled in the product trial period will show the study group as product trial in the listings when applicable.


Appendix 16.1.10.1 Clinical Laboratory Reference Ranges by Site

| Site | Laboratory Group | Test Name | Gender | Age Category | Normal Range | Unit |
|---|---|---|---|---|---|---|
| XXX | Serum Chemistry | Test Name | <i>⇔</i> | <> <> | XX - XX | units |
| | - | Test Name | $\Leftrightarrow$ | $\Leftrightarrow$ | XX - XX | units |
| | | Test Name | $\Leftrightarrow$ | $\Diamond$ | XX - XX | units |
| | Hematology | Test Name | <> | $\Leftrightarrow$ | XX - XX | units |
| | | Test Name | $\Leftrightarrow$ | $\Diamond$ | XX - XX | units |
| | | Test Name | $\Leftrightarrow$ | $\Diamond$ | XX - XX | units |
| | | Test Name | <> | $\Diamond$ | XX - XX | units |
| | | Test Name | $\Leftrightarrow$ | $\Diamond$ | XX - XX | units |

Note: Site XXX = <description of sites>

Program: /CAXXXXX/sas\_prg/stsas/lis\_PROGRAMNAME.sas DDMMMYYYY HH:MM

**Programmer Note: Similar for remaining Laboratory Groups and Test Names.** 

Appendix 16.2.1.1 Subject Disposition and Discontinuation (Randomized)

| Site | Subject<br>Number | Randomization<br>Number | Study<br>Group | Product<br>Assignment | Date | Completed<br>Study? | Day | Reason for<br>Discontinuation | Specify |
|---|---|---|---|---|---|---|---|---|---|
| XXX | XXXXXX | XXX | Х | X | DDMMYYYY | Yes | | | |
| | XXXXXX | XXX | X | X | DDMMYYYYY | Yes | | | |
| | XXXXXX | XXX | X | X | DDMMYYYYY | Yes | | | |
| | XXXXXX | XXX | X | X | DDMMYYYYY | Yes | | | |
| | XXXXXX | XXX | X | X | DDMMYYYYY | No | XXX | Personal Reason | |
| | XXXXXX | XXX | X | X | DDMMYYYY | Yes | | | |
| | XXXXXX | XXX | X | X | DDMMYYYYY | Yes | | | |
| | XXXXXX | XXX | X | X | DDMMYYYYY | Yes | | | |

Note: Group X = <description of groups>

Product A = Subject's OB Cigarette (Reference Product)

Product A = Subject's OB Cigarette (Reference Product)

Product B = Oral tobacco-derived nicotine chews marketed as VERVE® Discs Blue Mint (~1.5 mg nicotine/piece) (Test Product)

Product C = Oral tobacco-derived nicotine chews marketed as VERVE® Discs Green Mint (~1.5 mg nicotine/piece) (Test Product)

Product D = Oral tobacco-derived nicotine chews marketed as VERVE® Chews Blue Mint (~1.5 mg nicotine/piece) (Test Product)

Product E = Oral tobacco-derived nicotine chews marketed as VERVE® Chews Green Mint (~1.5 mg nicotine/piece) (Test Product)

Site XXX = <description of sites>

Appendix 16.2.1.2 Subject Disposition and Discontinuation (Product Trial)

| Site | Subject<br>Number | Discontinuation<br>Date | Day | Completed<br>Study? | Reason for<br>Discontinuation | Specify |
|---|---|---|---|---|---|---|
| XXX | XXXXXX | DDMMYYYY | X | <br>No | XXXXXXXXXXXX | |
| | XXXXXX | DD <b>MM</b> YYYY | X | No | XXXXXXXXXXX | |
| | XXXXXX | DD <b>MM</b> YYYY | X | No | XXXXXXXXXX | |
| | XXXXXX | DD <b>MM</b> YYYY | X | No | XXXXXXXXXXXX | |
| | XXXXXX | DD <b>MM</b> YYYY | X | No | XXXXXXXXXX | |

Note: Site XXX = <description of sites>

Appendix 16.2.1.3 Subject Disposition and Discontinuation (Screen Failures)

| Site | Subject<br>Number | Discontinuation<br>Date | Completed<br>Study? | Reason for<br>Discontinuation | Specify |
|---|---|---|---|---|---|
| XXX | XXXXXX | DDMMYYYY | No | XXXXXXXXXXXX | |
| | XXXXXX | DD <b>M</b> MYYYY | No | XXXXXXXXXXX | |
| | XXXXXX | DD <b>M</b> MYYYY | No | XXXXXXXXXX | |
| | XXXXXX | DD <b>M</b> MYYYY | No | XXXXXXXXXXXXX | |
| | XXXXXX | DDMMYYYY | No | XXXXXXXXX | |

Note: Site XXX = <description of sites>

Appendix 16.2.4.1.1 Demographics (I of II)

| Site | Subject<br>Number | Study<br>Group | Age<br>(yrs) | Gender | Race | Ethnicity | Reproductive<br>Status | Height<br>(cm) | Weight<br>(kg) | BMI<br>(kg/m^2) |
|---|---|---|---|---|---|---|---|---|---|---|
| XXX | XXXXXX | Х | XX | XXXX | XXXXXXXXX | XXXXXXXXXXX | XXXXXXXXXX | XX.X | XXX.X | XX.XX |
| | XXXXXX | X | XX | XXXX | XXXXXXXX | XXXXXXXXXXX | XXXXXXXXXX | XX.X | XXX.X | XX.XX |
| | XXXXXX | X | XX | XXXX | XXXXXXXXX | XXXXXXXXXXX | XXXXXXXXXX | XX.X | XXX.X | XX.XX |

Note: BMI = Body Mass Index

Group X = <description of groups>

Site XXX = <description of sites>

Appendix 16.2.4.1.2 Demographics (II of II)

| Site | Subject<br>Number | Study<br>Group | Informed<br>Consent<br>Date | Informed<br>Re-Consent<br>Date | Protocol<br>Version |
|---|---|---|---|---|---|
| XXX | XXXXXX | X | DDMMYYYY | DDMMYYYY | XXXXXXX |
| | XXXXXX | X | DDMMYYYY | DDMMYYYYY | XXXXXXX |
| | XXXXXX | X | DDMMYYYY | DDMMYYYYY | XXXXXXX |
| | XXXXXX | X | DDMMYYYY | DDMMYYYY | XXXXXXX |
| | XXXXXX | X | DDMMYYYY | DDMMYYYYY | XXXXXXX |
| | XXXXXX | X | DDMMYYYY | DDMMYYYYY | XXXXXXX |

Note: Group X = <description of groups>

Site XXX = <description of sites>

Appendix 16.2.4.1.3 Subject Characteristics

| Site | Subject<br>Number | Study<br>Group | Was Subject<br>Characteristics<br>Collected? | Date of<br>Collection | Annual<br>Household<br>Income | Highest Grade<br>or Year of School<br>Completed |
|---|---|---|---|---|---|---|
| XXX | XXXXXX | Х | XXX | DDMMYYYY | XXXXXXXXX | XXXXXXXXXXX |
| 2447 | | | | | XXXXXXXXXX | |
| | XXXXXX | X | XXX | DDMMYYYY | XXXXXXXXX | XXXXXXXXXXX |
| | XXXXXX | X | XXX | DDMMYYYY | XXXXXXXX | XXXXXXXXXX |
| | XXXXXX | X | XXX | DDMMYYYYY | XXXXXXXXX | XXXXXXXXXX |
| | XXXXXX | X | XXX | DDMMYYYYY | XXXXXXXXX | XXXXXXXXXX |
| | XXXXXX | X | XXX | DDMMYYYYY | XXXXXXXXX | XXXXXXXXXX |

Note: Group = <description of groups>

Site XXX = <description of sites>


#### Appendix 16.2.4.2.1 Physical Examination (I of II)

| | Visi | t | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Subject<br>Number | Name | Date | Day | Study<br>Group | | | Reason for<br>Not Done | System1 | System2 | System3 | System4 | System5 |
| XXXXXX | Screening | DDMMYYYY | | X | | XXX | | XXXXXXX | XXXXXXX | XXXXXXX | XXXXXXX | XXXXXXX |
| | XXXXXXX | DDMMYYYY | -X | | X | XXX | | XXXXXXX | XXXXXXX | XXXXXXX | XXXXXXX | XXXXXXX |
| | End of Study | DDMMYYYY | XX | | X | XXX | | XXXXXXX | XXXXXXX | XXXXXXX | XXXXXXX | XXXXXXX |

Note: See Appendix 16.2.4.2.3 for physical examination abnormality descriptions.

Group X = <description of groups>

### Appendix 16.2.4.2.2 Physical Examination (II of II)

| | Visi | t | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Subject<br>Number | Name | Date | Day | Study<br>Group Product | System6 | System7 | System8 | System9 | System10 | etc. |
| XXXXXX | Screening<br>XXXXXXXX<br>End of Study | DDMMYYYY<br>DDMMYYYYY<br>DDMMYYYYY | | X<br>X<br>X<br>X | XXXXXXX<br>XXXXXXX<br>XXXXXXX | XXXXXXX<br>XXXXXXX<br>XXXXXXX | XXXXXXX<br>XXXXXXX<br>XXXXXXX | XXXXXXX<br>XXXXXXX<br>XXXXXXX | XXXXXXX<br>XXXXXXX<br>XXXXXXX | XXXXXXX<br>XXXXXXX<br>XXXXXXX |

Note: See Appendix 16.2.4.2.3 for physical examination abnormality descriptions.

Group X = <description of groups>

### Appendix 16.2.4.2.3 Physical Examination Descriptions

| Visit<br>Subject | | | | | | Observatory | | | 0 | 011-1-11- |
|---|---|---|---|---|---|---|---|---|---|---|
| | Number | Name | Date | Day | Group | Study<br>Product | Result | System | Specify if Abnormal or Not Done | Significant? |
| | XXXXXX | Screening | DDMMYYYY | | X | | ABNORMAL | Skin | RIGHT CHEST SCAR | NCS |
| | XXXXXX | XXXXXX | DDMMYYYY | XX | Χ | X | ABNORMAL | Skin | ABDOMINAL SCAR | NCS |
| | XXXXXX | Screening | DDMMYYYY | | Х | | ABNORMAL | Skin | ABDOMINAL SCAR | NCS |

Note: NCS = Not clinically significant

Group X = <description of groups>


### Appendix 16.2.4.3 Medical History

| | | Visit | | | Date | | Were any | |
|---|---|---|---|---|---|---|---|---|
| Subject<br>Number | Any<br>History? | Name Date | History<br>Number | Report Term | Start | End | Ongoing? | comcomitant medications taken? |
| XXXXXX | XXX | Screening DDMMMYYYY | 1<br>2 | XXXXXX XXXXX<br>XXXXXX XXXXX | MMYYYY<br>MMYYYY | MMYYYY | YES<br>NO | XXX<br>XXX |
| XXXXXX | XXX | Screening DDMMMYYYY | 1 | XXXXXX XXXXX | MMYYYY | | YES | XXX |

Appendix 16.2.4.4.1 Tobacco/Nicotine Product Use History (I of II)

| Visit | | | | | | | | | | Cig | arette | Smoked | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Subject<br>Number | Name | Date | Study<br>Group | Not<br>Done? | Reason for<br>Not Done | | Quit? | Duration | Unit | CPD | Brand | Brand Style | Flavor | Length (mm) |
| XXXXXX | Screening | DDMMYYYY | X | | | XX | XXXX | XX | XXXX | XXX | XXXX | XXXX | XXXX | XX |
| XXXXXX | Screening | DDMMYYYYY | X | | | XX | XXXX | XX | XXXX | XXX | XXXX | XXXX | XXXX | XX |

Note: Group X = <description of groups>

Nicotine Replacement = Are you currently using a nicotine replacement therapy patch, gum, inhaler, nasal spray or lozenge? Quit? = Do you plan to quit smoking in the next 30 days? Duration = How long have you smoked cigarettes?

CPD = How many cigarettes do you typically smoke per day?

Appendix 16.2.4.4.2 Tobacco/Nicotine Product Use History (II of II)

| Subject<br>Number | | sit<br><br>Date | Study<br>Group | Tobacco Product | EVER Used<br>Even Once? | Used in the Past 30 days? |
|---|---|---|---|---|---|---|
| XXXXXX | Screening | DDMMMYYYY | X | XXXXXXXXXXXXXX<br>XXXXXXXXXXXXXXX<br>XXXXXXXX | XXX<br>XXX<br>XXX | XX<br>XX<br>XX<br>XX |

Note: Group X = <description of groups>

Appendix 16.2.4.5 Fagerström Test for Cigarette Dependence


| | Vi | .sit | | | Answer | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Subject<br>Number | Name | Date | Study<br>Group | Not<br>Done? Question 1 | Question 2 | Question 3 | Question 4 | Question 5 | Question 6 | FTCD<br>Score |
| XXXXXX | Screening | DDMMYYYY | X | XXXXXXXXX | XXX | XXXXXXXXXXX | XXXXXXXXXX | XXX | XXX | Χ |
| XXXXXX | Screening | DDMMYYYY | X | XXXXXXXX | XXX | XXXXXXXXXXX | XXXXXXXXX | XXX | XXX | X |
| XXXXXX | Screening | DDMMYYYYY | X | XXXXXXXXX | XXX | XXXXXXXXXXXX | XXXXXXXXXX | XXX | XXX | X |

Note: Question 1 = How soon after you wake up do you smoke your first cigarette?

Question 2 = Do you find it difficult to refrain from smoking in places where it is forbidden, e.g., in church, at the library,

cinema, etc?

Question 3 = Which cigarette would you hate most to give up?

Question 4 = How many cigarettes/day do you smoke?

Question 5 = Do you smoke more frequently during the first hours of waking than during the rest of the day?

Question 6 = Do you smoke if you are so ill that you are in bed most of the day?

Group X = <description of groups>


### Appendix 16.2.5.1 Inclusion / Exclusion Criteria Not Met

| Curlo di o o t | Visit | | Met All Study Eligibility | | Inclusion/ | C | |
|---|---|---|---|---|---|---|---|
| Subject<br>Number | Name | Date | Group | Criteria? | Exclusion<br>Category | Criterion<br>Identifier | Criterion |
| | _ | DDMMYYYY<br>DDMMYYYYY | | Yes<br>No | XX | xxxx | ×××××××××××××××××××××××××××××××××××××× |

Note: Group X = <description of groups>


### Appendix 16.2.5.2.1 Product Trial

| Subject<br>Number | Visit | Study<br>Group | | oject Willing<br>Verve products? | VERVE Product | Date | Start<br>Time | Stop<br>Time |
|---|---|---|---|---|---|---|---|---|
| XXXXXX | XXXXX | Х | X | XXX | xxxxxxxxx | DDMMYYY | HH:MM | HH:MM |

Note: Group X = <description of groups>

#### Appendix 16.2.5.2.2 In-Clinic Product Use

| Subject | Study | Study | Episode | Product | Dispense | Dispense | Product | Return | Returned | Comment |
|---|---|---|---|---|---|---|---|---|---|---|
| Number | Day | Group | # | Dispense | Date | Time | Returned? | Date | Time | |
| XXXXXX | XXXXX | | 1 | XXX | DDMMMYYY | HH:MM | XXX | DDMMYYYY | HH:MM | |

Note: Group X = <description of groups>

Appendix 16.2.5.2.3 Max CPD

| Subject<br>Number | | 2 | Max CPD<br>Not Done | Reason for<br>Not Done | Maximum CPD<br>Allowed |
|---|---|---|---|---|---|
| XXXXXX | XXXXX | × | XX | XXX | XX |

Note: Group X = <description of groups>

Appendix 16.2.5.3.1 24-Hour Urine Collection


| Subjec | t Study | Study | Planned | Was Collection | | | | _ | | | Incomplete, | | , |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| _ | | | | Performed? | | Time | | | _ | | discarded | | Specify |
| XXXXXX | Х | X | XXXXX | XXX | <br>DDMMYYYY | HH:MM | DDMMYYYYY | HH:MM | XXXX | XX | XXX | XXX | |

Note: Group X = <description of groups>

Product X = <description of products>

Appendix 16.2.5.3.2 Urine Samples


| Subject Study<br>Number Group | 4 | | <u> </u> | Creatinine- Samples Collected (2 aliquots of 5mL each) | Exposure (2 aliquots | 2 | Biobanking<br>(2 aliquots<br>of 40mL each) |
|---|---|---|---|---|---|---|---|
| XXXXXX X | X | XXXXX | X | X | X | X | X |

Note: Group X = <description of groups>

Product X = <description of products>


### Appendix 16.2.5.4 Carboxyhemoglobin Blood Collection

| | | | | | Colle | ection | |
|---|---|---|---|---|---|---|---|
| Subject | Study | Study | Planned | Was Blood Sample | | | How Many COHb Samples |
| Number | Group | Product | Timepoint | for COHb collected? | Date | Time | Were Collected? |
| XXXXXX | X | X | XXXXX | XXX | DD <b>MM</b> YYYY | HH:MM | X |

Note: Group X = <description of groups>

Product X = <description of products>


### Appendix 16.2.5.5 Prior and Concomitant Medications

| | | | | Medication/<br>? Therapy | | Dosage | Route | | Start<br>Time | I | Stop<br>Time | Frequency | Indication | Continuing? | AE# |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| XXXXXX | Х | X | XXX | ACETAMINOPHE | EN XX | 620 mg | ORAL | DDMMY | YYYY HH:MM | DDMMYYY | Y HH: | MM Once | Toothache | e No | XXX |

Note: Group X = <description of groups>

Product X = <description of products>

Appendices 16.2.6.1 through 16.2.6.18 will have the following format:

Appendix 16.2.6.1 Total Urine NNAL


| Subject<br>Number | Study<br>Group | Study<br>Product | | | Urine<br>Weight<br>(g) | Mass | Absolute Change<br>From Baseline<br>(unit) | % Change From<br>Baseline | Creatinine<br>Conc.<br>(mg/dL) | Adjusted for<br>Urine Creatinine<br>(mass/g Cr) |
|---|---|---|---|---|---|---|---|---|---|---|
| XXXXX | Х | X | -1<br>5<br>7 | XXX<br>XXX<br>XXX | XXX<br>XXX<br>XXX | XXX<br>XXX<br>XXX | NA<br>XXX<br>XXX | NA<br>XXX<br>XXX | XXX<br>XXX<br>XXX | XXX<br>XXX<br>XXX<br>XXX |

Note: Baseline = Day -1, Conc. = Concentration

Group X = <description of groups>

Product X = <description of products>


### Appendix 16.2.6.3.1 Urine Nicotine and Metabolites Concentrations

| Subject<br>Number | Study<br>Group | Study<br>product | Study<br>Day | Nicotine<br>(ng/mL) | Nicotine<br>Glucuronide<br>(ng/mL) | Cotinine<br>(ng/mL) | Cotinine<br>Glucuronide<br>(ng/mL) | Trans-3-hydroxy<br>Cotinine<br>(ng/mL) | Trans-3-nydroxy<br>Cotinine<br>Glucuronide<br>(ng/mL) | |
|---|---|---|---|---|---|---|---|---|---|---|
| XXXXXX | X | X | - <u>1</u> | XXX<br>XXX | XXX | XXX | XXXX | XXX | XXX | _ |
| | | | 7 | XXX | XXX<br>XXX | XXX<br>XXX | XXXX | XXX<br>XXX | XXX<br>XXX | |

Note: Group X = <description of groups>

Product X = <description of products>

#### Appendix 16.2.6.19 Blood COHb

| Subject<br>Number | | | | | Absolute Change<br>From Baseline<br>(unit) | % Change From<br>Baseline |
|---|---|---|---|---|---|---|
| XXXXX | Х | Х | -1<br>5<br>7 | XXX<br>XXX<br>XXX | NA<br>XXX<br>XXX | NA<br>XXX<br>XXX |

Note: Baseline = Day -1, Conc. = Concentration

Group X = <description of groups>

Product X = <description of products>

Appendix 16.2.6.20.1 Cigarettes Used per Day

| Subject<br>Number | | | | Cigarettes | Per Day |
|---|---|---|---|---|---|
| xxxxx | Х | Х | -2<br>-1<br>Baseline<br>1<br>2<br>3<br>4<br>5<br>6 | XX | |

Note: Baseline = Average of Days -2 and -1.

Group X = <description of groups>

Product X = <description of products>

Appendix 16.2.6.20.2 VERVE Product Used per Day

| Subject<br>Number | Study<br>Group | Study<br>Product | Study<br>Day | VERVE Product Used per Da | ıy |
|---|---|---|---|---|---|
| XXXXX | Х | Х | 1<br>2<br>3<br>4<br>5<br>6<br>7 | XX<br>XX<br>XX<br>XX<br>XX<br>XX<br>XX | |

Note: Group X = <description of groups>

Product X = <description of products>

Appendix 16.2.6.21.1 Duration of VERVE Product Used per Use

| Subject | Study | Study | Study | Episode | Duration |
|---|---|---|---|---|---|
| Number | Group | Product | Day | Number | (min) |
| XXXXX | X | X | 1 | 1<br>2<br>3 | XX.X<br>XX.X<br>XX.X<br>XX.X |

Note: Group X = <description of groups>

Product X = <description of products>

Appendix 16.2.6.21.2 Total Duration of VERVE Product Used per Day

| Subject<br>Number | Study<br>Group | Study<br>Product | Study<br>Day | Total Duration (min) |
|---|---|---|---|---|
| XXXXX | Х | Х | 1<br>2<br>3<br>4<br>5<br>6<br>7 | XX.X<br>XX.X<br>XX.X<br>XX.X<br>XX.X<br>XX.X<br>XX.X |

Note: Group X = <description of groups>

Product X = <description of products>

Appendix 16.2.6.22 Original and Factor Score to QSU-Brief Questionnaire

| | | | | | | | | | | | QST | J–Br: | lef | | | | Factor | Score |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Subject<br>Number | Study<br>Group | Study<br>Product | Study<br>Day | Time<br>Point | Date | Time | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 1 | 2 |
| XXXXX | X | X | -1 | Morning | DDMMYYYY | HH:MM:SS | Х | Х | X | Х | Х | Х | Х | Х | Х | Χ | X | X |
| | | | | Evening | DDMMYYYYY | HH:MM:SS | X | X | X | X | X | X | X | X | X | X | X | X |
| | | | | Change - | DDMMYYYY | | X | X | X | X | X | X | X | X | X | X | X | X |

Note: 1. I have a desire for a cigarette right now. 2. Nothing would be better than smoking a cigarette right now.

- 3. If it were possible, I would probably smoke right now.
- 4. I could control things better right now if I could smoke.
- 5. All I want right now is a cigarette. 6. I have an urge for a cigarette.
- 7. A cigarette would taste good right now. 8. I would do almost anything for a cigarette right now.
- 9. Smoking would make me less depressed. 10. I am going to smoke as soon as possible.

Factor Score 1 (anticipation of pleasure from smoking) = Average of items 1, 3, 6, 7, and 10

Facore Score 2 (relief of nicotine withdrawal) = Average of items 2, 4, 5, 8, and 9.

Change = Evening score - Morning score

Group X = <description of groups>

Product X = <description of products>

Appendix 16.2.6.23.1 Original Score to MCEQ Questionnaire

| 0.1. | Q1 1 | G1 1 | Q1 1 | | | | | | | | ľ | nCEQ | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Subject<br>Number | Group | Study<br>Product | Study<br>Day | Questionnaire | Date | Time | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 |
| XXXXX | X | Х | -1 | mCEQ-C | DDMMYYYY | HH:MM:SS | X | Х | X | X | X | X | X | X | X | X | X | X |
| | | | 1 | mCEQ-C | DDMMYYYYY | HH:MM:SS | X | X | X | X | X | X | X | X | Χ | X | X | X |
| | | | | mCEQ-V | DDMMYYYY | HH:MM:SS | X | X | X | Χ | X | X | X | X | Χ | X | X | X |
| | | | 5 | mCEQ-C | DDMMYYYY | HH:MM:SS | X | X | X | X | X | X | X | X | X | X | X | X |
| | | | | mCEO-V | DDMMMYYYY | HH:MM:SS | X | X | X | X | X | X | X | X | X | X | X | X |

Note: 1. Was using the product satisfying? 2. Did the product taste good?

- 3. Did you enjoy the sensations in your throat and chest? 4. Did using the product calm you down?
- 5. Did using the product make you feel more awake? 6. Did using the product make you feel less irritable?
- 7. Did using the product help you concentrate? 8. Did using the product reduce your hunger for food? 9. Did using the product make you dizzy? 10. Did using the product make you nauseous?
- 11. Did using the product immediately relieve your craving for a cigarette? 12. Did you enjoy using the product?

Group X = <description of groups>

Product X = <description of products>

Appendix 16.2.6.23.2 Factor Score to MCEQ Questionnaire


| Subject<br>Number | Study<br>Group | Study<br>Product | Study<br>Day | Questionnaire | Date | Time | Smoking<br>Satisfaction | Psychologica<br>Reward | Aversion | Enjoyment o<br>Sensation | of Craving<br>Reduction |
|---|---|---|---|---|---|---|---|---|---|---|---|
| XXXXX | X | X | -1 | mCEQ-C | DDMMYYYY | HH:MM:SS | X | X | X | X | X |
| | | | 1 | mCEQ-C | DDMMYYYYY | HH:MM:SS | X | X | X | X | X |
| | | | | mCEQ-V | DDMMYYYYY | HH:MM:SS | X | X | X | X | X |
| | | | 5 | mCEQ-C | DDMMYYYYY | HH:MM:SS | X | X | X | X | X |
| | | | | mCEO-V | DDMMMYYYY | HH·MM·SS | × | X | X | X | × |

Note: Smoking satisfaction: average of 1,2,12;

Psychological reward: average of 4 to 8; Aversion: average of 9,10;

Aversion: average of 9,10; Enjoyment of sensation: 3; Craving Reduction: 11

Group X = <description of groups>

Product X = <description of products>

Appendix 16.2.6.24 Use the Product Again Questionnaire


| Subject<br>Number | | Study<br>Product | Study<br>Day | Date | Time | If Given the Opportunity, I Would<br>Want to Use the Cigarette Again (mm) | Category | Bipolar<br>score |
|---|---|---|---|---|---|---|---|---|
| XXXXX | X | Х<br>Х | 7<br>7 | DDMMYYYY<br>DDMMMYYYY | | | -50 to <0<br>>0 to 50 | -XX<br>XX |

Note: Group X = <description of groups>

Product X = <description of products>

#### Appendix 16.2.7.1 Adverse Events (I of II)

Time from


| Ordo do o o | C+ | O+ | | 7.17 | | | Last<br>Product Use | Onset | | Resolve | d | Duration |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Subject<br>Number | Group | Study<br>Product | UE?^ | AE<br>Numbei | r Adverse Event* | Preferred Term | (DD:HH:MM) | Date | Time | Date | Time | (DD:HH:MM) |
| <br>XXXXXX | X | X | XXX | XX | XXXXXXXXXXX | XXXXXXXXX XXXXXX | XX:XX:XX | DDMMYYYY | HH:MM | DDMMYYYY | HH:MM | XX:XX:XX |
| XXXXXX | Χ | X | XXX | XX | XXXXXXXXXXX | XXXXXXXXX XXXXXXX | XX:XX:XX | DDMMYYYY | HH:MM | DDMMYYYY | HH:MM | XX:XX:XX |
| XXXXXX | X | X | XXX | XX | XXXXXXXXXXX | XXXXXXXXX XXXXXXX | XX:XX:XX | DDMMYYYY | HH:MM | DDMMYYYY | HH:MM | XX:XX:XX |
| XXXXXX | X | X | XXX | XX | XXXXXXXXXXX | XXXXXXXXX XXXXXXX | XX:XX:XX | DDMMYYYY | HH:MM | DDMMYYYY | HH:MM | XX:XX:XX |

Note: ^ UE = study product use-emergent \* = Adverse events are classified according to the MedDRA Version 20.0.

Group X = <description of groups>

Product X = <description of products>

Appendix 16.2.7.2 Adverse Events (II of II)


| Subje | act Stud | ly Study | Æ | Adverse | Onset | | | | | | Relationship to | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Numbe | er Grou | ip Product | | | Date | Time | Frequency | Severity | Serious | Outcome | Study Product | Action |
| XXXXX | X X | X | XX | XXXXXXXXX | DDMMYYYY | HH:MM | XXXXXXX | XXXXX | XXXX | XXXXXX | XXXXXXXX | XXXXX |
| XXXXX | X X | X | XX | XXXXXXXXX | DDMMYYYY | HH:MM | XXXXXXX | XXXXX | XXXX | XXXXXX | XXXXXXX | XXXXX |
| XXXXX | X X | X | XX | XXXXXXXXX | DDMMYYYY | HH:MM | XXXXXXX | XXXXX | XXXX | XXXXXX | XXXXXXX | XXXXX |
| XXXXX | X X | Х | XX | XXXXXXXXXX | DDMMYYYY | HH:MM | XXXXXXX | XXXXX | XXXX | XXXXXX | XXXXXXX | XXXXX |

Note: Group X = <description of groups>

Product X = <description of products>

Appendix 16.2.7.3 Adverse Event Preferred Term Classification

| Cl | C+ | C+ | 7.17 | 7 | | | | Onse | et. |
|---|---|---|---|---|---|---|---|---|---|
| Number | Group | Product | AE<br>Number | Adverse<br>Event | | Preferred Term | Body System | Date | Time |
| XXXXXX | X | X | XX | XXXXXXX | XXXXX XXXX XXXXXX | XXXXXXXXX XXXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | DDMMYYYY | HH:MM |
| XXXXXX | X | X | XX | XXXXXXX I | XXXXX XXXX XXXXXX | XXXXXXXXX XXXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | DDMMYYYY | HH:MM |
| XXXXXX | Χ | X | XX | XXXXXXX | XXXXX XXXX XXXXXX | XXXXXXXXX XXXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | DDMMYYYY | HH:MM |
| XXXXXX | Х | Х | XX | XXXXXXX I | XXXXX XXXX XXXXXX | XXXXXXXXXX XXXXXXX | *************************************** | DDMMYYYY | HH:MM |

Note: \* = Adverse events are classified according to the MedDRA Version 20.0.

Group X = <description of groups>

Product X = <description of products>

Program: /CAXXXXX/sas prg/stsas/lis PROGRAMNAME.sas DDMMYYYYY HH:MM


Appendices 16.2.8.1.2 to 16.2.8.1.3 will have the following format.

Page 1 of X Appendix 16.2.8.1.1 Clinical Laboratory Report - Serum Chemistry

| Subject | Age/ | Study Study | Visi | t<br> | | Parameter1 | Parameter2 | Parameter3 | Parameter4 | Parameter5 |
|---|---|---|---|---|---|---|---|---|---|---|
| Site Number | | Group Product | Name | Date | Date | | | | | |
| XXX XXXXXX | XX/X | X<br>X | Screening<br>XXXXXX | DDMMYYYY<br>DDMMYYYYY | | | XX<br>XX | XX<br>XX<br>XX | XX<br>XX | XX HN<br>XX HN |

Note: Refer to Appendix 16.1.10.1 for the reference ranges of clinical laboratory tests. H = Above Reference Range, L = Below Reference Range PI Interpretation: N = Not Clinically Significant

Group  $X = \langle description \ of \ groups \rangle$ 

Product X = <description of products>

Program: /CAXXXXX/sas prg/stsas/lis PROGRAMNAME.sas DDMMMYYYY HH:MM

Programmer Note: Replace Parameter1, 2 etc. with actual lab tests in the study.

Appendix 16.2.8.1.4 Clinical Laboratory Report - Comments


| Subject<br>Number | Study<br>Group | Study<br>Product | Visit | Date | Department | Test | Result | Unit | Comment |
|---|---|---|---|---|---|---|---|---|---|
| XXXXXX | X | X | XXXXXXX | DDMMYYYY | Other Tests | XXXXXXXX | XXX | mg/dL | Not significant in the |

Note: Group X = <description of groups>

Product X = <description of products>


Appendix 16.2.8.1.5 Alcohol Breath Tests

| Subject | Study | Visi | t<br> | Was an Alcohol<br>Breath Test | Test | |
|---|---|---|---|---|---|---|
| Number | Group | Name | Date | Performed? | Date | Result |
| XXXXXX | X | Screening<br>Check-in | DDMMYYYY<br>DDMMYYYY | XXX<br>XXX | DDMMYYYY<br>DDMMYYYY | XXXXXX<br>XXXXXX |

Note: Group X = <description of groups>


Appendix 16.2.8.1.6 Urine Drug Screens

| | | Visit | | | | | |
|---|---|---|---|---|---|---|---|
| Subject<br>Number | | Name | Date | Was the Urine<br>Sample Collected? | Date of<br>Collection | Test Name | Result |
| XXXXXX | Χ | Screening | DDMMYYYY | XXX | DDMMYYYY | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXXXXX |

Note: Group X = <description of groups>

Appendix 16.2.8.1.7 Pregnancy Tests


| Visit | | | Was the | | Collection | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Subject<br>Number | Study<br>Group | Name | Date | - Pregnancy<br>Test Done? | Reason for<br>Not Done | Date | Time | Category | Test<br>Name | Test<br>Result | Test<br>Code |
| XXXXXX | <u>-</u> | <br>Screening | DDMMYYYY | XXX | | DDMMYYYY | HH:MM | XXXXXX | XXXX | XXX | XXXX |
| | | XXXXXXXXX | DDMMYYYYY | XXX | | DDMMYYYYY | HH:MM | XXXXXX | XXXX | XXX | XXXX |

Note: Group X = <description of groups>

Appendix 16.2.8.1.8 Serum FSH


| | | Vis | sit | Was Serum | | | |
|---|---|---|---|---|---|---|---|
| Subject | Study | | | FSH | Reason for | Was Postmenopausal | Collection |
| Number | Group - | Name | Date | Done? | Not Done | Status confirmed? | Date |
| | | | DD1000000000 | | | 1777 | DD10000000 |
| XXXXXX | X | Screening | DDMMYYYY | XXX | | XXX | DDMMYYYYY |

Note: Group X = <description of groups>

Appendix 16.2.8.1.9 Contraception


| Subject | Study - | Vis | it<br> | | | Double | Intrauterine | Vasectomized | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Number | Group | Name | Date | Contraception | on? Hormonal | Barrier? | Device? | Partner? | Other | Specify |
| XXXXXX | X | Screening | DDMMYYYY<br>DDMMYYYYY | XXX | XXX | XXX | XXX | XXX | | |

Note: Group X = <description of groups>

Appendix 16.2.8.1.10 Urine Cotinine Screens


| Subject<br>Number | | Visi<br>Name | t<br>Date | Was the Urine<br>Cotinine Sample<br>Collected? | | Result (ng/mL) |
|---|---|---|---|---|---|---|
| XXXXXX | Χ | Screening | DDMMYYYY | XXX | DDMMYYYY | XXX |

Note: Group X = <description of groups>


Appendix 16.2.8.1.11 Serology Sample Collection

| | | Vis | it | | Collection |
|---|---|---|---|---|---|
| Subject<br>Number | Study<br>Group | Name | Date | Was the Sample<br>Collected? | Date |
| XXXXXX | X | Screening | DDMMYYYYY | XXX | DDMMYYYY |

Note: Group X = <description of groups>

#### Appendix 16.2.8.2 Vital Signs


| Subject<br>Number | Name | Study<br>Group | Study<br>Product | Date | Time | Not<br>Done? | Reasor<br>Not<br>Done | n Blood Pressure (mmHg<br><br>Systolic/Diastolic | - Pulse | Respi-<br>ration<br>(rpm) | Tempe-<br>rapture<br>(°F) |
|---|---|---|---|---|---|---|---|---|---|---|---|
| XXXXXX | Screening<br>Check-in<br>End-of-Study | X | X | DDMMYYYY<br>DDMMYYYYY<br>DDMMMYYYY | HH:MM<br>HH:MM<br>HH:MM | | | XXX/ XX<br>XXX/ XX NCS<br>XXX/ XX | XX<br>XX<br>XX CS | XX<br>XX<br>XX | XX.X<br>XX.X<br>XX.X |

Note: NCS = Not clinically significant, CS = Clinically significant

Group X = <description of groups>

Product X = <description of products>

Appendix 16.2.8.3 12-Lead Electrocardiogram


| | | | | | | Heart | | | | | If Abi | normal |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Subject | | Study | | | | Rate | PR | QRS | QΤ | QTcB* | | |
| Number | Visit | Group | Date | Time | Result | (bpm) | (ms) | (ms) | (ms) | (ms) | Specify | Action Taken |
| XXXXXX | Screeni | ng X | DDMMMYYYY | HH:MM | Normal | XX | XXX | XX | XXX | XXX | | |

Note: QTCB\* = QTc corrected using Bazett's correction, ANCS = Abnormal, Not Clinically Significant

Group X = <description of groups>


Appendix 16.2.8.4 Smoking Cessation Information

| Subject | Visit | Was Smoking Cessation | Date<br>Information |
|---|---|---|---|
| Subject<br>Number | Visit | Was Smoking Cessation<br>Information Offered? | Offered |
| XXXXXX | Screening<br>End of Study | XXX<br>XXX | DDMMYYYY<br>DDMMYYYY |

## 14. FIGURE SHELLS

Box plots will be presented as in the figure below, with the headings of Baseline, Visit 5 or Visit 7:

Figure 14.2.4.1.1
Box Plot of Total Urine NNAL at Baseline and Day 7 by Study Group (mITT Population)



The upper and lower whiskers of the boxplot represent, respectively, the largest and smallest observed values within 1.5 × the interquartile range (IQR) from the upper and lower quartiles (Q3 and Q1). Values greater or smaller than the bounds represented by these whiskers are identified as extreme values with the corresponding subject number.

Program: CAXXXXX/XXX PROGRAMNAME.SAS DDMMMYYYY HH:MM

#### 15. REFERENCES

- 1. Sanderson L et al. 2001. Evaluation of the brief questionnaire of smoking urges (QSU-brief) in laboratory and clinical settings. Nicotine and Tobacco Research. (3)7-16
- 2. Cappelleri et al. 2007. Confirmatory factor analysis and reliability of the modified cigarette evaluation questionnaire. Additive Behaviors. (32)912-923.